CLINICAL TRIAL: NCT03287310
Title: A Randomised Double-blind (Sponsor Open), Placebo Controlled, Single Ascending Dose, First Time in Human Study in Participants With Mild to Moderate Asthma to Assess Safety, Tolerability, Immunogenicity, Pharmacokinetics and Pharmacodynamics of GSK3511294 Administered Subcutaneously
Brief Title: First Time in Human (FTIH) Study to Evaluate Safety, Tolerability, Immunogenicity, Pharmacokinetics (PK) and Pharmacodynamics (PD) of GSK3511294 Administered Subcutaneously (SC) in Subjects With Mild to Moderate Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205722; 2016-004256-30 (EudraCT Number)
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Results first posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Asthma
Keywords: eosinophils; pharmacokinetics; First time in Human; GSK3511294; pharmacodynamics; asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Intervention Model Description: This is a multi-center, double-blind study in which subjects will be allocated to five cohorts. The subjects in each cohort will be randomized to receive GSK3511294 and placebo in a ratio of 3:1. In each cohort, dosing will be staggered: one subject will receive GSK3511294 and one subject will receive placebo at least 72 hours before the remaining subjects in that cohort are dosed. The remaining subjects will be dosed if the review of all safety data up to 72 hours after dosing of the first two subjects in each cohort is satisfactory.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Subjects receiving GSK3511294 in Cohort 1 (Experimental): Six subjects in Cohort 1 will receive a single SC dose of 2 mg GSK3511294.
  Interventions: Drug: GSK3511294; Drug: Salbutamol/albuterol
- Subjects receiving placebo in Cohort 1 (Placebo Comparator): Two subjects in Cohort 1 will receive a single SC dose of placebo.
  Interventions: Drug: Placebo; Drug: Salbutamol/albuterol
- Subjects receiving GSK3511294 in Cohort 2 (Experimental): Six subjects in Cohort 2 will receive a single SC dose of 10 mg GSK3511294.
  Interventions: Drug: GSK3511294; Drug: Salbutamol/albuterol
- Subjects receiving placebo in Cohort 2 (Placebo Comparator): Two subjects in Cohort 2 will receive a single SC dose of placebo.
  Interventions: Drug: Placebo; Drug: Salbutamol/albuterol
- Subjects receiving GSK3511294 in Cohort 3 (Experimental): Nine subjects in Cohort 3 will receive a single SC dose of 30 mg GSK3511294.
  Interventions: Drug: GSK3511294; Drug: Salbutamol/albuterol
- Subjects receiving placebo in Cohort 3 (Placebo Comparator): Three subjects in Cohort 3 will receive a single SC dose of placebo.
  Interventions: Drug: Placebo; Drug: Salbutamol/albuterol
- Subjects receiving GSK3511294 in Cohort 4 (Experimental): Nine subjects in Cohort 4 will receive a single SC dose of 100 mg GSK3511294.
  Interventions: Drug: GSK3511294; Drug: Salbutamol/albuterol
- Subjects receiving placebo in Cohort 4 (Placebo Comparator): Three subjects in Cohort 4 will receive a single SC dose of placebo.
  Interventions: Drug: Placebo; Drug: Salbutamol/albuterol
- Subjects receiving GSK3511294 in Cohort 5 (Experimental): Six subjects in Cohort 5 will receive a single SC dose of 300 mg GSK3511294.
  Interventions: Drug: GSK3511294; Drug: Salbutamol/albuterol
- Subjects receiving placebo in Cohort 5 (Placebo Comparator): Two subjects in Cohort 5 will receive a single SC dose of placebo.
  Interventions: Drug: Placebo; Drug: Salbutamol/albuterol

INTERVENTIONS:
Drug: GSK3511294 — GSK3511294 will be available as a clear or opalescent, colorless or yellow to brown solution for injection at unit dose strength of 150 milligrams per milliliter (mg/mL). GSK3511294 will be diluted in 0.9% weight by volume (w/v) sodium chloride to achieve the desired concentration for administration. GSK3511294 will be administered by SC injection.
  Arms: Subjects receiving GSK3511294 in Cohort 1; Subjects receiving GSK3511294 in Cohort 2; Subjects receiving GSK3511294 in Cohort 3; Subjects receiving GSK3511294 in Cohort 4; Subjects receiving GSK3511294 in Cohort 5
Drug: Placebo — Matching Placebo will consist of 0.9% w/v sodium chloride which will be administered by the SC route.
  Arms: Subjects receiving placebo in Cohort 1; Subjects receiving placebo in Cohort 2; Subjects receiving placebo in Cohort 3; Subjects receiving placebo in Cohort 4; Subjects receiving placebo in Cohort 5
Drug: Salbutamol/albuterol — Salbutamol/albuterol will be supplied to all subjects for use as rescue medication during the study.

SUMMARY:
GSK3511294 is a humanized monoclonal antibody antagonist of Interleukin (IL)-5 which is known to block binding of IL-5 to the IL-5 receptor complex, causing a reduction in the circulating population of eosinophils. This is a single ascending dose FTIH study to investigate safety, tolerability, immunogenicity, pharmacokinetics (PK) and pharmacodynamics (PD) of GSK3511294, administered SC in subjects with mild to moderate asthma maintained on a low-medium daily dose of inhaled corticosteroids (ICS) or ICS/long acting beta-agonist (LABA), and short acting beta-agonist (SABA). The subjects will attend a pre-screen visit of up to 12 weeks before dosing for assessment of blood eosinophils. Eligible subjects with blood eosinophils >=200 cells per microliter (cells/µL) will undergo a screening period of up to 4 weeks. The subjects will then be randomized into 5 cohorts. In each cohort, the subjects will be randomized to receive a single dose of GSK3511294 or placebo in a ratio of 3:1. The follow-up period will be up to 40 weeks post dose and will be dose-dependent. The scheduled maximum duration for each subject will be up to 44 weeks including up to 28 days of screening.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should be between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Blood eosinophils of >= 200 cells/µL at screening.
* A physician diagnosis of asthma (mild or moderate, as defined by the Global Initiative for Asthma [GINA], 2017) at least 12 months prior to the start of the study. The reason for diagnosis of asthma should be documented in the subject's source data, including relevant history and investigations - specifically evidence of airway hyper-responsiveness, airflow variation (peak flow rate or forced expiratory volume in one second [FEV1]) or reversible airflow obstruction should also be documented in the subject's source data.
* A screening pre-bronchodilator FEV1 >= 60% of predicted normal value.
* Asthma Control Test score > 19.
* hsCRP of < 10 milligrams per liter (mg/L) at screening.
* Otherwise healthy (other than the acceptable conditions of asthma and other atopic diseases, including allergic rhinitis and atopic dermatitis) based on a screening medical history, physical examination, vital signs, ECG assessment, pulmonary function testing, and clinical laboratory results.
* Maintained controlled on as needed SABA and one of the following: a) stable dose of ICS; b) stable dose of combination therapy: ICS/LABA.
* Body weight >= 50 kilograms (kg), and body mass index (BMI) of 19-32 kilograms per square meter (kg/m^2) inclusive.
* Male and female subjects. a) a female subject is eligible to participate if she is not pregnant, not breastfeeding, and not a woman of childbearing potential. b) as GSK3511294 is a monoclonal antibody that is not anticipated to interact directly with Deoxyribonucleic acid (DNA) or other chromosomal material with minimal exposure through semen expected, male subjects will not be required to use contraception during the study, nor are they prohibited from donating sperm.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions of the study.

Exclusion Criteria:

* Any asthma exacerbation requiring systemic corticosteroids within 12 weeks of screening, or that resulted in overnight hospitalization requiring additional treatment for asthma within 6 months prior to screening.
* A history of life-threatening asthma defined as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest or hypoxic seizures within the last 5 years.
* Significant pulmonary diseases, other than asthma, including (but not limited to): pneumonia previously requiring hospital admission, pulmonary fibrosis, bronchopulmonary dysplasia, chronic bronchitis, emphysema, chronic obstructive pulmonary disease, or other significant respiratory abnormalities.
* Suspected or confirmed bacterial or viral infection (including tuberculosis) of the upper or lower respiratory tract, sinus or middle ear that occurred within and/or has not resolved within 4 weeks of screening that: led to a change in asthma management or in the opinion of the Investigator, is expected to affect the subject's asthma status or the subject's ability to participate in the study.
* Positive for hepatitis B surface antigen (HBsAg) at screening.
* Positive hepatitis C antibody test result at screening, or within 3 months prior to first dose of study treatment.
* Known immunodeficiency (other than that explained by the use of corticosteroids), including a positive test for human immunodeficiency virus (HIV) antibody at screening.
* Latent or chronic infections (example, genital herpes, urinary tract infections) or at risk of infection (example, significant trauma or infection within the 90 days before screening).
* Opportunistic infection within 6 months prior to screening (example, a non-tuberculous mycobacterial infection or cytomegalovirus, pneumocystosis, aspergillosis).
* Parasitic infestation within 6 months prior to screening, or have travelled to a country with a high prevalence of such infections in the 6 months before screening, or intend to do so in the year after dosing.
* Live vaccine within 4 weeks prior to screening, or intention to receive live vaccine during the study.
* Corrected QT by Fridericia's formula (QTcF) interval > 450 milliseconds (msec)
* A personal history of severe hypertension, arrhythmia, Right Bundle Branch Block, or Left Bundle Branch Block, or a family history of sudden unexplained death, long QT, familial cardiac syndrome, or cardiomyopathy.
* ALT >1.5 times upper limit of normal (ULN).
* Bilirubin >1.5 times ULN. Isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Any history or presence of clinically relevant cardiac or cardiovascular, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, or infectious disease or immunodeficiency, or signs of acute illness, or any other illness or condition that, in the opinion of the investigator (in consultation with the medical monitor), would adversely affect the subject's participation in this study.
* A previous history of cancer in remission for less than 5 years prior to screening (except for localized carcinoma of the skin that had been resected for cure) or current malignancy.
* A positive drug/alcohol test before dosing, OR any history of drug abuse OR regular alcohol consumption within 6 months of the study defined as: An average weekly intake of > 14 units alcohol. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (equivalent to 240 milliliters [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Current smokers or ex-smokers who have given up smoking for < 12 months and/or have a smoking pack history of > 5 pack years (1 pack year = 20 cigarettes per day for 1 year or 5 cigarettes per day for 4 years).
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Anticipated non-availability and/or risk of non-compliance with study visits and procedures, or unwillingness or inability to follow the study specific procedures.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 3 months, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first dosing day.
* History of sensitivity to any of the study medications, or its components, or a history of drug reaction or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Major surgery within 90 days prior to screening, or planned in-patient surgery or hospitalization during the study period
* Donation or loss of blood or blood products in excess of 500 mL within the 3 months before dosing.
* History of renal disease, abnormal kidney function or evidence of persisting or clinically relevant protein or blood on urinalysis.
* History or signs of immunologically active disease (including the presence of low C3 or low C4) or thrombocytopenia.
* History of vasculitis.
* Subjects are excluded if they are undergoing desensitization therapy, or have received any of the following medications as indicated prior to screening: anti- Immunoglobulin E (IgE) therapy (within 6 months); anti-IL5 (within 6 months); oral or injectable corticosteroids (within 8 weeks); long acting muscarinic antagonist (LAMA) or leukotriene receptor antagonist (LTRA) therapy (within 8 weeks); drugs that can prolong the QT interval.
* Subjects who are employees of the sponsor or clinical unit are excluded.
* Vulnerable subjects, e.g., participants kept in detention, protected adults under guardianship, trusteeship and soldiers, or participants committed to an institution by governmental or juridical order.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Germany (2):
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Berlin
- United Kingdom (3):
  - GSK Investigational Site, Harrow, Middlesex
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request Site
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Singh D, Fuhr R, Bird NP, Mole S, Hardes K, Man YL, Cahn A, Yancey SW, Pouliquen IJ. A Phase 1 study of the long-acting anti-IL-5 monoclonal antibody GSK3511294 in patients with asthma. Br J Clin Pharmacol. 2022 Feb;88(2):702-712. doi: 10.1111/bcp.15002. Epub 2021 Aug 24. PMID 34292606

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was double-blind, placebo-controlled, single ascending dose study in participants with mild to moderate asthma to assess safety, tolerability, immunogenicity, pharmacokinetics and pharmcodynamics of GSK3511294 administered subcutaneously. The study was conducted in Germany and United Kingdom.
Pre-assignment Details: A total of 50 participants were enrolled in this study, of which two did not receive any study treatment and 48 were included in the Safety Population.
Groups:
- Placebo: Participants were administered a single subcutaneous dose of GSK3511294 matching placebo on Day 1
- GSK3511294 2 mg: Participants were administered a single subcutaneous dose of GSK3511294 2 milligram (mg) on Day 1
- GSK3511294 10 mg: Participants were administered a single subcutaneous dose of GSK3511294 10 mg on Day 1
- GSK3511294 30 mg: Participants were administered a single subcutaneous dose of GSK3511294 30 mg on Day 1
- GSK3511294 100 mg: Participants were administered a single subcutaneous dose of GSK3511294 100 mg on Day 1
- GSK3511294 300 mg: Participants were administered a single subcutaneous dose of GSK3511294 300 mg on Day 1
Period: Overall Study
Arm/Group | Placebo | GSK3511294 2 mg | GSK3511294 10 mg | GSK3511294 30 mg | GSK3511294 100 mg | GSK3511294 300 mg
Started | 12 | 6 | 6 | 9 | 9 | 6
Completed | 12 | 6 | 6 | 9 | 9 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- GSK3511294 2mg: Participants were administered a single subcutaneous dose of GSK3511294 2 milligram (mg) on Day 1
- GSK3511294 10mg: Participants were administered a single subcutaneous dose of GSK3511294 10 mg on Day 1
- GSK3511294 30mg: Participants were administered a single subcutaneous dose of GSK3511294 30 mg on Day 1
- GSK3511294 100mg: Participants were administered a single subcutaneous dose of GSK3511294 100 mg on Day 1
- GSK3511294 300mg: Participants were administered a single subcutaneous dose of GSK3511294 300 mg on Day 1
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg | Total
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (13.37) | 43.5 (10.71) | 44.7 (13.20) | 44.9 (10.23) | 42.0 (10.84) | 45.2 (11.18) | 44.0 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Male | 12 | 6 | 6 | 9 | 8 | 5 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Central/South Asian Heritage | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Black or African American (Afr. Amer.) | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Arabic/North African Heritage | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White/Caucasian/European Heritage | 9 | 5 | 6 | 7 | 9 | 6 | 42
  Black/Afr. Amer./White/Caucasian/European Heritage | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs (SAE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; other important medical events that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed before; is associated with liver injury and impaired liver function.
Time Frame: Up to Week 40
Population: Safety Population comprised of all randomized participants who received at least one dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Participants
  Any AE | 11 | 2 | 6 | 8 | 9 | 4
  Any SAE | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Adverse Events of Special Interest (AESI)
Description: AESIs were defined as Hypersensitivity (narrow) and Injection site reactions like hematoma and swelling.
Time Frame: Up to Week 40
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Participants
  Hypersensitivity | 0 | 0 | 0 | 1 | 0 | 0
  Injection Site Reaction: hematoma | 1 | 0 | 0 | 0 | 0 | 1
  Injection Site Reaction: swelling | 1 | 0 | 0 | 0 | 0 | 1

3. Primary Outcome: Change From Baseline in Neutrophil, Lymphocyte, Monocyte, Eosinophil, Basophil and Platelet Count
Description: Blood samples were collected at indicated time-points for analysis of hematology parameters like platelet count, neutrophils, lymphocytes, monocytes, eosinophils and basophils. Baseline was defined as latest pre-dose assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 2, 3, 4 and 5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32, 36 and 40
Population: Safety Population. Only those participants with planned assessments at that particular time point has been presented (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Giga cells per liter
  Basophils, Day 2,n=12,6,6,8,9,6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 9 | 6
  Basophils, Day 2,n=12,6,6,8,9,6 | -0.006 (0.0247) | -0.020 (0.0297) | 0.003 (0.0103) | -0.003 (0.0238) | 0.001 (0.0302) | -0.018 (0.0160)
  Basophils, Day 3,n=12,6,6,9,9,6 | 0.002 (0.0356) | 0.003 (0.0450) | 0.010 (0.0126) | -0.003 (0.0260) | -0.003 (0.0224) | -0.007 (0.0121)
  Basophils, Day 4,n=12,6,6,8,8,6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 8 | 6
  Basophils, Day 4,n=12,6,6,8,8,6 | -0.003 (0.0296) | 0.002 (0.0214) | -0.008 (0.0325) | -0.004 (0.0207) | -0.001 (0.0136) | 0.002 (0.0214)
  Basophils, Day 5,n=11,6,6,9,9,6: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 6
  Basophils, Day 5,n=11,6,6,9,9,6 | -0.020 (0.0224) | -0.008 (0.0204) | -0.020 (0.0141) | -0.009 (0.0196) | -0.003 (0.0255) | -0.025 (0.0164)
  Basophils, Week 1,n=12,6,6,9,9,5: number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 5
  Basophils, Week 1,n=12,6,6,9,9,5 | -0.001 (0.0257) | -0.017 (0.0207) | -0.018 (0.0306) | 0.002 (0.0291) | 0.001 (0.0162) | -0.006 (0.0055)
  Basophils, Week 2,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Basophils, Week 2,n=12,6,5,9,9,6 | -0.006 (0.0215) | -0.018 (0.0204) | 0.000 (0.0274) | -0.004 (0.0224) | -0.007 (0.0158) | -0.007 (0.0137)
  Basophils, Week 4,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Basophils, Week 4,n=12,6,5,9,9,6 | -0.010 (0.0316) | -0.002 (0.0232) | -0.004 (0.0167) | 0.002 (0.0172) | -0.006 (0.0265) | -0.010 (0.0126)
  Basophils, Week 8,n=12,6,6,9,9,6 | 0.005 (0.0183) | 0.007 (0.0266) | -0.022 (0.0271) | -0.010 (0.0122) | -0.002 (0.0186) | -0.015 (0.0138)
  Basophils, Week 12,n=12,5,6,9,9,5: number analyzed (Participants) | 12 | 5 | 6 | 9 | 9 | 5
  Basophils, Week 12,n=12,5,6,9,9,5 | 0.002 (0.0229) | -0.014 (0.0297) | -0.008 (0.0147) | -0.003 (0.0245) | -0.004 (0.0142) | -0.006 (0.0055)
  Basophils, Week 18,n=12,6,6,9,9,6 | -0.002 (0.0229) | 0.010 (0.0310) | -0.012 (0.0160) | -0.001 (0.0267) | 0.010 (0.0278) | -0.005 (0.0105)
  Basophils, Week 24,n=11,6,6,9,9,6: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 6
  Basophils, Week 24,n=11,6,6,9,9,6 | -0.005 (0.0157) | 0.002 (0.0264) | -0.005 (0.0288) | -0.004 (0.0313) | -0.001 (0.0154) | -0.018 (0.0117)
  Basophils, Week 26,n=12,6,6,9,9,6 | -0.004 (0.0284) | 0.002 (0.0306) | 0.000 (0.0219) | 0.008 (0.0383) | -0.002 (0.0199) | -0.008 (0.0133)
  Basophils, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Basophils, Week 32,n=6,6,6,0,0,6 | -0.002 (0.0376) | 0.010 (0.0210) | 0.005 (0.0339) |  |  | -0.008 (0.0117)
  Basophils, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Basophils, Week 36,n=6,0,0,9,9,0 | -0.002 (0.0214) |  |  | 0.021 (0.0247) | -0.002 (0.0199) |
  Basophils, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Basophils, Week 40,n=2,0,0,0,0,6 | 0.000 (0.0000) |  |  |  |  | -0.012 (0.0313)
  Eosinophils, Day 2,n=12,6,6,8,9,6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 9 | 6
  Eosinophils, Day 2,n=12,6,6,8,9,6 | 0.024 (0.1412) | -0.120 (0.0587) | -0.145 (0.0797) | -0.251 (0.1504) | -0.208 (0.1685) | -0.152 (0.0794)
  Eosinophils, Day 3,n=12,6,6,9,9,6 | -0.001 (0.1986) | -0.167 (0.0755) | -0.203 (0.0876) | -0.289 (0.0987) | -0.287 (0.1744) | -0.182 (0.0920)
  Eosinophils, Day 4,n=12,6,6,8,8,6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 8 | 6
  Eosinophils, Day 4,n=12,6,6,8,8,6 | 0.014 (0.1950) | -0.172 (0.0749) | -0.212 (0.1144) | -0.348 (0.1149) | -0.300 (0.1829) | -0.192 (0.0643)
  Eosinophils, Day 5,n=11,6,6,9,9,6: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 6
  Eosinophils, Day 5,n=11,6,6,9,9,6 | -0.034 (0.1529) | -0.202 (0.0799) | -0.235 (0.1117) | -0.326 (0.1385) | -0.276 (0.1351) | -0.210 (0.0767)
  Eosinophils, Week 1,n=12,6,6,9,9,5: number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 5
  Eosinophils, Week 1,n=12,6,6,9,9,5 | 0.033 (0.1461) | -0.195 (0.0609) | -0.242 (0.1189) | -0.324 (0.1350) | -0.298 (0.1824) | -0.206 (0.0568)
  Eosinophils, Week 2,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Eosinophils, Week 2,n=12,6,5,9,9,6 | 0.072 (0.1809) | -0.212 (0.0895) | -0.210 (0.0886) | -0.344 (0.1334) | -0.307 (0.1602) | -0.223 (0.0952)
  Eosinophils, Week 4,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Eosinophils, Week 4,n=12,6,5,9,9,6 | 0.025 (0.1635) | -0.227 (0.0712) | -0.238 (0.1150) | -0.366 (0.1466) | -0.321 (0.1969) | -0.253 (0.0855)
  Eosinophils, Week 8,n=12,6,6,9,9,6 | 0.036 (0.1486) | -0.230 (0.0769) | -0.280 (0.1202) | -0.379 (0.1519) | -0.343 (0.1841) | -0.252 (0.1007)
  Eosinophils, Week 12,n=12,5,6,9,9,5: number analyzed (Participants) | 12 | 5 | 6 | 9 | 9 | 5
  Eosinophils, Week 12,n=12,5,6,9,9,5 | 0.025 (0.1566) | -0.174 (0.0777) | -0.262 (0.1087) | -0.371 (0.1484) | -0.336 (0.1895) | -0.250 (0.1245)
  Eosinophils, Week 18,n=12,6,6,9,9,6 | 0.029 (0.1263) | -0.148 (0.0685) | -0.208 (0.1153) | -0.359 (0.1445) | -0.338 (0.1786) | -0.253 (0.1067)
  Eosinophils, Week 24,n=11,6,6,9,9,6: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 6
  Eosinophils, Week 24,n=11,6,6,9,9,6 | -0.021 (0.1436) | -0.072 (0.0662) | -0.103 (0.1916) | -0.300 (0.1546) | -0.334 (0.1769) | -0.245 (0.1017)
  Eosinophils, Week 26,n=12,6,6,9,9,6 | 0.035 (0.1812) | -0.042 (0.0571) | -0.037 (0.2813) | -0.273 (0.1773) | -0.319 (0.1724) | -0.252 (0.0920)
  Eosinophils, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Eosinophils, Week 32,n=6,6,6,0,0,6 | 0.008 (0.0935) | 0.042 (0.1153) | 0.003 (0.2467) |  |  | -0.235 (0.1205)
  Eosinophils, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Eosinophils, Week 36,n=6,0,0,9,9,0 | -0.045 (0.1758) |  |  | -0.041 (0.2734) | -0.258 (0.1594) |
  Eosinophils, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Eosinophils, Week 40,n=2,0,0,0,0,6 | 0.245 (0.1344) |  |  |  |  | -0.222 (0.1196)
  Lymphocytes, Day 2,n=12,6,6,8,9,6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 9 | 6
  Lymphocytes, Day 2,n=12,6,6,8,9,6 | -0.010 (0.3897) | 0.135 (0.2886) | 0.108 (0.2185) | -0.061 (0.3165) | -0.157 (0.3336) | 0.100 (0.2804)
  Lymphocytes, Day 3,n=12,6,6,9,9,6 | 0.064 (0.4447) | 0.330 (0.3571) | 0.143 (0.1810) | -0.140 (0.2382) | -0.081 (0.4131) | 0.143 (0.3296)
  Lymphocytes, Day 4,n=12,6,6,8,8,6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 8 | 6
  Lymphocytes, Day 4,n=12,6,6,8,8,6 | 0.006 (0.4963) | 0.193 (0.3242) | 0.172 (0.3474) | 0.005 (0.1753) | 0.005 (0.3798) | 0.210 (0.2772)
  Lymphocytes, Day 5,n=11,6,6,9,9,6: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 6
  Lymphocytes, Day 5,n=11,6,6,9,9,6 | -0.077 (0.4746) | 0.108 (0.2319) | 0.085 (0.1302) | -0.253 (0.2983) | 0.104 (0.4463) | 0.047 (0.1226)
  Lymphocytes, Week 1,n=12,6,6,9,9,5: number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 5
  Lymphocytes, Week 1,n=12,6,6,9,9,5 | 0.048 (0.4628) | 0.295 (0.2404) | 0.058 (0.4116) | -0.060 (0.3248) | -0.018 (0.4217) | -0.154 (0.2587)
  Lymphocytes, Week 2,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Lymphocytes, Week 2,n=12,6,5,9,9,6 | -0.133 (0.4107) | 0.222 (0.3543) | 0.096 (0.4117) | -0.120 (0.3304) | -0.068 (0.4104) | 0.047 (0.1189)
  Lymphocytes, Week 4,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Lymphocytes, Week 4,n=12,6,5,9,9,6 | -0.189 (0.4616) | 0.088 (0.2938) | 0.056 (0.2899) | -0.062 (0.2346) | -0.052 (0.5189) | -0.137 (0.2103)
  Lymphocytes, Week 8,n=12,6,6,9,9,6 | -0.057 (0.4665) | 0.105 (0.2670) | -0.107 (0.3584) | -0.188 (0.2277) | 0.052 (0.3287) | -0.075 (0.0672)
  Lymphocytes, Week 12,n=12,5,6,9,9,5: number analyzed (Participants) | 12 | 5 | 6 | 9 | 9 | 5
  Lymphocytes, Week 12,n=12,5,6,9,9,5 | -0.142 (0.4107) | 0.228 (0.1968) | 0.072 (0.4113) | 0.014 (0.2490) | 0.048 (0.3231) | -0.388 (0.2237)
  Lymphocytes, Week 18,n=12,6,6,9,9,6 | -0.212 (0.4094) | -0.032 (0.2213) | -0.042 (0.3612) | -0.097 (0.4088) | 0.050 (0.4539) | -0.063 (0.1788)
  Lymphocytes, Week 24,n=11,6,6,9,9,6: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 6
  Lymphocytes, Week 24,n=11,6,6,9,9,6 | -0.179 (0.3876) | -0.028 (0.3616) | -0.040 (0.2744) | -0.070 (0.3102) | 0.052 (0.9838) | -0.132 (0.1619)
  Lymphocytes, Week 26,n=12,6,6,9,9,6 | -0.088 (0.4361) | -0.223 (0.3808) | -0.138 (0.3577) | -0.116 (0.4946) | 0.018 (0.5392) | -0.188 (0.2566)
  Lymphocytes, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Lymphocytes, Week 32,n=6,6,6,0,0,6 | -0.165 (0.6851) | -0.057 (0.2842) | -0.197 (0.5467) |  |  | -0.148 (0.2017)
  Lymphocytes, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Lymphocytes, Week 36,n=6,0,0,9,9,0 | 0.007 (0.1838) |  |  | -0.043 (0.4393) | 0.006 (0.4176) |
  Lymphocytes, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Lymphocytes, Week 40,n=2,0,0,0,0,6 | 0.285 (0.3465) |  |  |  |  | -0.125 (0.2966)
  Monocytes, Day 2,n=12,6,6,8,9,6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 9 | 6
  Monocytes, Day 2,n=12,6,6,8,9,6 | -0.002 (0.0914) | 0.017 (0.1357) | 0.123 (0.1240) | 0.015 (0.1176) | 0.019 (0.0715) | 0.052 (0.1947)
  Monocytes, Day 3,n=12,6,6,9,9,6 | 0.029 (0.1001) | 0.028 (0.1533) | 0.100 (0.1235) | -0.028 (0.0753) | 0.032 (0.0952) | 0.018 (0.1514)
  Monocytes, Day 4,n=12,6,6,8,8,6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 8 | 6
  Monocytes, Day 4,n=12,6,6,8,8,6 | 0.032 (0.0936) | -0.002 (0.1258) | 0.118 (0.1057) | -0.038 (0.0927) | 0.068 (0.1074) | 0.050 (0.0434)
  Monocytes, Day 5,n=11,6,6,9,9,6: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 6
  Monocytes, Day 5,n=11,6,6,9,9,6 | -0.034 (0.0841) | -0.025 (0.0701) | 0.053 (0.1299) | -0.100 (0.1470) | 0.074 (0.1874) | -0.035 (0.0766)
  Monocytes, Week 1,n=12,6,6,9,9,5: number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 5
  Monocytes, Week 1,n=12,6,6,9,9,5 | 0.006 (0.0998) | 0.072 (0.1127) | 0.057 (0.1786) | 0.032 (0.0578) | 0.101 (0.1039) | -0.012 (0.0926)
  Monocytes, Week 2,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Monocytes, Week 2,n=12,6,5,9,9,6 | 0.013 (0.0945) | 0.050 (0.1621) | 0.056 (0.0451) | 0.004 (0.0975) | 0.118 (0.1738) | 0.090 (0.2697)
  Monocytes, Week 4,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Monocytes, Week 4,n=12,6,5,9,9,6 | 0.001 (0.0757) | 0.103 (0.1382) | -0.018 (0.0817) | 0.042 (0.0559) | 0.041 (0.1014) | -0.003 (0.1201)
  Monocytes, Week 8,n=12,6,6,9,9,6 | 0.048 (0.1377) | 0.123 (0.1681) | -0.053 (0.0484) | -0.006 (0.0648) | 0.080 (0.1211) | 0.058 (0.1509)
  Monocytes, Week 12,n=12,5,6,9,9,5: number analyzed (Participants) | 12 | 5 | 6 | 9 | 9 | 5
  Monocytes, Week 12,n=12,5,6,9,9,5 | 0.007 (0.1042) | 0.050 (0.0561) | -0.013 (0.0841) | 0.059 (0.0864) | 0.140 (0.1734) | 0.084 (0.1680)
  Monocytes, Week 18,n=12,6,6,9,9,6 | 0.042 (0.0897) | -0.040 (0.1362) | -0.045 (0.0944) | 0.018 (0.1475) | 0.092 (0.0874) | 0.043 (0.1516)
  Monocytes, Week 24,n=11,6,6,9,9,6: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 6
  Monocytes, Week 24,n=11,6,6,9,9,6 | 0.028 (0.1181) | -0.013 (0.0989) | 0.070 (0.0921) | 0.047 (0.1301) | 0.159 (0.2567) | 0.037 (0.0975)
  Monocytes, Week 26,n=12,6,6,9,9,6 | 0.040 (0.0888) | -0.037 (0.1129) | 0.010 (0.0551) | 0.036 (0.1267) | 0.121 (0.1500) | 0.013 (0.0720)
  Monocytes, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Monocytes, Week 32,n=6,6,6,0,0,6 | -0.035 (0.0817) | -0.013 (0.1600) | 0.098 (0.0783) |  |  | -0.012 (0.0662)
  Monocytes, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Monocytes, Week 36,n=6,0,0,9,9,0 | 0.067 (0.0717) |  |  | 0.053 (0.1624) | 0.158 (0.2126) |
  Monocytes, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Monocytes, Week 40,n=2,0,0,0,0,6 | 0.040 (0.0566) |  |  |  |  | -0.032 (0.0873)
  Platelet, Day 2,n=12,5,5,9,9,6: number analyzed (Participants) | 12 | 5 | 5 | 9 | 9 | 6
  Platelet, Day 2,n=12,5,5,9,9,6 | -9.7 (19.00) | -6.8 (10.40) | -6.4 (15.27) | -6.8 (17.99) | 6.1 (22.05) | -1.5 (19.32)
  Platelet, Day 3,n=12,5,6,9,9,6: number analyzed (Participants) | 12 | 5 | 6 | 9 | 9 | 6
  Platelet, Day 3,n=12,5,6,9,9,6 | -2.8 (16.72) | -9.4 (8.29) | 5.7 (13.00) | -7.1 (19.98) | 1.7 (19.24) | -0.8 (19.60)
  Platelet, Day 4,n=12,5,5,8,8,6: number analyzed (Participants) | 12 | 5 | 5 | 8 | 8 | 6
  Platelet, Day 4,n=12,5,5,8,8,6 | -5.6 (18.64) | -5.8 (3.63) | 6.6 (15.66) | -0.4 (18.86) | -1.1 (21.56) | -0.2 (6.62)
  Platelet, Day 5,n=12,5,6,9,9,6: number analyzed (Participants) | 12 | 5 | 6 | 9 | 9 | 6
  Platelet, Day 5,n=12,5,6,9,9,6 | -7.6 (17.59) | -3.6 (13.89) | -3.0 (18.11) | -4.6 (19.09) | 6.2 (22.90) | -2.8 (18.62)
  Platelet, Week 1,n=12,5,6,9,8,6: number analyzed (Participants) | 12 | 5 | 6 | 9 | 8 | 6
  Platelet, Week 1,n=12,5,6,9,8,6 | -0.9 (20.21) | -10.2 (11.30) | 5.0 (21.08) | -3.9 (12.41) | 16.8 (25.37) | -13.8 (28.69)
  Platelet, Week 2,n=12,5,6,9,9,6: number analyzed (Participants) | 12 | 5 | 6 | 9 | 9 | 6
  Platelet, Week 2,n=12,5,6,9,9,6 | 3.5 (16.51) | 2.8 (13.59) | -6.3 (29.38) | -0.9 (25.09) | 25.0 (38.64) | -15.5 (39.81)
  Platelet, Week 4,n=12,5,4,9,9,6: number analyzed (Participants) | 12 | 5 | 4 | 9 | 9 | 6
  Platelet, Week 4,n=12,5,4,9,9,6 | -11.5 (26.10) | -6.8 (20.93) | 1.3 (37.07) | -1.6 (17.61) | 12.3 (35.87) | -5.0 (22.80)
  Platelet, Week 8,n=12,5,5,9,9,6: number analyzed (Participants) | 12 | 5 | 5 | 9 | 9 | 6
  Platelet, Week 8,n=12,5,5,9,9,6 | 4.3 (22.85) | 11.6 (23.71) | 2.6 (29.01) | -11.3 (21.03) | 22.0 (30.81) | -3.5 (23.89)
  Platelet, Week 12,n=12,5,6,9,9,5: number analyzed (Participants) | 12 | 5 | 6 | 9 | 9 | 5
  Platelet, Week 12,n=12,5,6,9,9,5 | -14.8 (26.42) | -6.0 (16.63) | -9.0 (26.83) | -10.8 (10.15) | 27.4 (43.23) | -25.6 (24.39)
  Platelet, Week 18,n=12,5,6,9,9,6: number analyzed (Participants) | 12 | 5 | 6 | 9 | 9 | 6
  Platelet, Week 18,n=12,5,6,9,9,6 | -8.6 (21.65) | -13.4 (20.42) | -14.0 (9.53) | 1.6 (19.51) | 15.9 (22.45) | 2.2 (28.92)
  Platelet, Week 24,n=10,5,6,9,9,6: number analyzed (Participants) | 10 | 5 | 6 | 9 | 9 | 6
  Platelet, Week 24,n=10,5,6,9,9,6 | -1.9 (14.81) | -7.8 (18.35) | -10.0 (14.97) | -1.6 (19.94) | 19.7 (30.07) | -5.7 (39.38)
  Platelet, Week 26,n=12,5,6,9,9,6: number analyzed (Participants) | 12 | 5 | 6 | 9 | 9 | 6
  Platelet, Week 26,n=12,5,6,9,9,6 | 2.4 (30.14) | -13.8 (17.70) | -19.3 (13.81) | -2.4 (12.21) | 11.8 (36.37) | -6.8 (17.38)
  Platelet, Week 32,n=6,5,6,0,0,6: number analyzed (Participants) | 6 | 5 | 6 | 0 | 0 | 6
  Platelet, Week 32,n=6,5,6,0,0,6 | 5.5 (18.71) | -0.6 (15.37) | -6.3 (10.39) |  |  | -15.7 (51.15)
  Platelet, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Platelet, Week 36,n=6,0,0,9,9,0 | -1.8 (25.65) |  |  | -0.3 (12.37) | 13.9 (24.15) |
  Platelet, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Platelet, Week 40,n=2,0,0,0,0,6 | -20.0 (2.83) |  |  |  |  | -11.7 (30.80)
  Neutrophil, Day 2,n=12,6,6,8,9,6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 9 | 6
  Neutrophil, Day 2,n=12,6,6,8,9,6 | -0.078 (0.8813) | 0.413 (0.6493) | -0.005 (0.9228) | 0.301 (0.5042) | 0.241 (0.8219) | 0.102 (0.4630)
  Neutrophil, Day 3,n=12,6,6,9,9,6 | 0.161 (0.4542) | 0.015 (0.6691) | 0.225 (0.6850) | 0.077 (0.9525) | 0.217 (1.1014) | 0.038 (0.5158)
  Neutrophil, Day 4,n=12,6,6,8,8,6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 8 | 6
  Neutrophil, Day 4,n=12,6,6,8,8,6 | 0.390 (0.4832) | 0.560 (0.4666) | 0.438 (0.9293) | 0.151 (0.9472) | 0.130 (1.0414) | 0.215 (0.4194)
  Neutrophil, Day 5,n=11,6,6,9,9,6: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 6
  Neutrophil, Day 5,n=11,6,6,9,9,6 | 0.155 (0.7789) | 0.085 (0.6109) | -0.003 (0.3494) | 0.041 (0.7075) | 0.184 (1.0809) | 0.103 (0.2639)
  Neutrophil, Week 1,n=12,6,6,9,9,5: number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 5
  Neutrophil, Week 1,n=12,6,6,9,9,5 | -0.179 (0.6365) | -0.483 (1.2069) | -0.160 (0.3280) | -0.151 (0.5955) | 0.174 (0.8992) | 0.070 (0.4346)
  Neutrophil, Week 2,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Neutrophil, Week 2,n=12,6,5,9,9,6 | -0.209 (0.4662) | -0.738 (0.7110) | -0.142 (1.0604) | -0.192 (0.9481) | 0.229 (0.8853) | -0.310 (0.6362)
  Neutrophil, Week 4,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Neutrophil, Week 4,n=12,6,5,9,9,6 | -0.540 (0.4797) | -0.768 (0.7810) | -0.156 (0.9674) | -0.279 (0.5859) | -0.340 (0.7049) | 0.023 (0.7539)
  Neutrophil, Week 8,n=12,6,6,9,9,6 | -0.218 (0.7893) | 0.497 (1.6165) | -0.277 (0.9128) | -0.069 (1.0047) | -0.127 (0.5829) | 0.258 (0.5218)
  Neutrophil, Week 12,n=12,5,6,9,9,5: number analyzed (Participants) | 12 | 5 | 6 | 9 | 9 | 5
  Neutrophil, Week 12,n=12,5,6,9,9,5 | 0.043 (0.9639) | -0.712 (0.5890) | 0.053 (1.0187) | -0.180 (0.4760) | -0.344 (0.4840) | -0.362 (0.5607)
  Neutrophil, Week 18,n=12,6,6,9,9,6 | -0.093 (0.9727) | -0.158 (0.7786) | 0.015 (0.7474) | -0.012 (0.8076) | -0.151 (0.5728) | -0.027 (0.6629)
  Neutrophil, Week 24,n=11,6,6,9,9,6: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 6
  Neutrophil, Week 24,n=11,6,6,9,9,6 | -0.326 (0.4501) | -0.752 (0.9422) | -0.370 (0.3746) | -0.144 (0.5243) | 0.140 (0.5795) | -0.128 (0.4311)
  Neutrophil, Week 26,n=12,6,6,9,9,6 | -0.105 (0.7933) | -0.527 (0.6332) | -0.622 (0.6065) | -0.259 (0.9389) | 0.104 (0.7127) | -0.295 (0.2855)
  Neutrophil, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Neutrophil, Week 32,n=6,6,6,0,0,6 | -0.393 (0.8219) | -0.708 (0.7757) | 0.880 (1.9211) |  |  | -0.360 (0.3275)
  Neutrophil, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Neutrophil, Week 36,n=6,0,0,9,9,0 | -0.163 (0.8441) |  |  | -0.384 (0.4763) | -0.004 (0.9080) |
  Neutrophil, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Neutrophil, Week 40,n=2,0,0,0,0,6 | -0.005 (0.1061) |  |  |  |  | 0.332 (0.3452)

4. Primary Outcome: Change From Baseline in Red Blood Cell Count (RBC)
Description: Blood samples were collected at indicated time-points for analysis of hematology parameters like RBC count. Baseline was defined as latest pre-dose assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 2, 3, 4 and 5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32, 36 and 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Trillion cells per liter
  Day 2,n=12,6,6,9,9,6 | -0.08 (0.212) | -0.07 (0.197) | 0.08 (0.223) | 0.00 (0.194) | 0.16 (0.246) | 0.05 (0.243)
  Day 3,n=12,6,6,9,9,6 | 0.03 (0.214) | -0.08 (0.133) | 0.13 (0.242) | 0.01 (0.190) | 0.06 (0.133) | 0.03 (0.186)
  Day 4,n=12,6,6,8,8,6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 8 | 6
  Day 4,n=12,6,6,8,8,6 | -0.04 (0.211) | -0.08 (0.133) | 0.10 (0.179) | -0.03 (0.149) | 0.04 (0.185) | 0.10 (0.141)
  Day 5,n=12,6,6,9,9,6 | -0.18 (0.175) | -0.22 (0.133) | -0.10 (0.261) | -0.08 (0.120) | 0.03 (0.316) | 0.05 (0.187)
  Week 1,n=12,6,6,9,9,5: number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 5
  Week 1,n=12,6,6,9,9,5 | -0.15 (0.215) | -0.37 (0.175) | 0.00 (0.190) | -0.03 (0.218) | 0.07 (0.180) | -0.02 (0.147)
  Week 2,n=12,6,6,9,9,6 | -0.11 (0.156) | -0.28 (0.133) | -0.18 (0.183) | -0.07 (0.206) | 0.11 (0.232) | -0.08 (0.194)
  Week 4,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Week 4,n=12,6,5,9,9,6 | -0.18 (0.248) | -0.35 (0.055) | -0.16 (0.230) | -0.08 (0.192) | 0.09 (0.293) | -0.03 (0.137)
  Week 8,n=12,6,6,9,9,6 | -0.03 (0.253) | -0.23 (0.186) | -0.02 (0.248) | -0.13 (0.200) | 0.18 (0.277) | 0.07 (0.103)
  Week 12,n=12,6,6,9,9,5: number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 5
  Week 12,n=12,6,6,9,9,5 | -0.13 (0.176) | -0.25 (0.138) | -0.05 (0.251) | -0.01 (0.237) | 0.19 (0.237) | 0.00 (0.141)
  Week 18,n=12,6,6,9,9,6 | -0.02 (0.292) | -0.20 (0.219) | -0.08 (0.271) | -0.02 (0.228) | 0.27 (0.283) | 0.17 (0.163)
  Week 24,n=11,6,6,9,9,6: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 6
  Week 24,n=11,6,6,9,9,6 | -0.11 (0.221) | -0.27 (0.175) | -0.05 (0.164) | 0.01 (0.169) | 0.13 (0.229) | 0.17 (0.151)
  Week 26,n=12,6,6,9,9,6 | -0.12 (0.301) | -0.33 (0.216) | -0.08 (0.204) | -0.02 (0.120) | 0.20 (0.194) | 0.12 (0.117)
  Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Week 32,n=6,6,6,0,0,6 | -0.10 (0.237) | -0.18 (0.183) | 0.08 (0.248) |  |  | 0.05 (0.176)
  Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Week 36,n=6,0,0,9,9,0 | 0.12 (0.232) |  |  | 0.10 (0.122) | 0.33 (0.357) |
  Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Week 40,n=2,0,0,0,0,6 | -0.05 (0.071) |  |  |  |  | 0.12 (0.098)

5. Primary Outcome: Change From Baseline in Mean Corpuscle Volume (MCV)
Description: Blood samples were collected at indicated time-points for analysis of hematology parameters like MCV. Baseline was defined as latest pre-dose assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 2, 3, 4 and 5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32, 36 and 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Femtoliters
  Day 2,n=12,6,6,9,9,6 | 0.2 (0.94) | 0.2 (0.75) | 0.2 (0.75) | 0.1 (2.85) | -0.3 (1.00) | 1.3 (2.16)
  Day 3,n=12,6,6,9,9,6 | 0.7 (1.07) | -0.3 (0.82) | 0.2 (0.75) | 0.0 (1.32) | -1.0 (1.41) | 0.3 (1.37)
  Day 4,n=12,6,6,8,8,6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 8 | 6
  Day 4,n=12,6,6,8,8,6 | 0.3 (0.78) | -0.5 (1.05) | 0.0 (1.26) | -0.1 (0.83) | -1.8 (0.89) | 0.2 (0.98)
  Day 5,n=12,6,6,9,9,6 | 1.3 (1.92) | 0.5 (0.55) | 0.3 (0.82) | 2.0 (2.92) | -1.0 (3.50) | 0.7 (1.75)
  Week 1,n=12,6,6,9,9,6 | -0.2 (0.94) | -0.8 (1.33) | 0.2 (0.75) | -1.2 (1.20) | -1.7 (2.06) | -0.7 (1.21)
  Week 2,n=12,6,6,9,9,6 | 0.0 (1.28) | -0.3 (1.51) | 0.2 (0.75) | -0.9 (1.17) | -1.4 (2.51) | -0.3 (1.63)
  Week 4,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Week 4,n=12,6,5,9,9,6 | 0.7 (2.39) | -0.8 (2.14) | 0.2 (0.45) | -0.7 (0.87) | -1.6 (2.13) | -0.2 (0.98)
  Week 8,n=12,6,6,9,9,6 | 0.3 (1.23) | -0.3 (1.51) | 0.2 (0.75) | 0.0 (1.12) | -2.2 (2.91) | -0.2 (1.17)
  Week 12,n=12,6,6,9,9,5: number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 5
  Week 12,n=12,6,6,9,9,5 | 0.5 (1.09) | -1.2 (1.94) | 0.2 (0.75) | -0.7 (1.87) | -2.4 (2.55) | -1.2 (0.84)
  Week 18,n=12,6,6,9,9,6 | -0.4 (1.73) | -0.8 (1.33) | 0.5 (1.64) | -1.9 (1.05) | -2.8 (3.07) | -1.0 (1.10)
  Week 24,n=11,6,6,9,9,6: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 6
  Week 24,n=11,6,6,9,9,6 | -0.8 (1.78) | -0.3 (1.86) | 0.8 (1.72) | -1.6 (1.51) | -2.4 (3.54) | -0.7 (1.03)
  Week 26,n=12,6,6,9,9,6 | -0.5 (2.24) | 0.0 (2.10) | 0.5 (0.84) | -1.7 (1.58) | -2.3 (3.04) | -0.3 (1.03)
  Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Week 32,n=6,6,6,0,0,6 | 0.5 (1.38) | 0.0 (2.45) | 0.8 (1.47) |  |  | -0.2 (0.98)
  Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Week 36,n=6,0,0,9,9,0 | -1.5 (1.05) |  |  | -1.9 (1.05) | -1.8 (2.44) |
  Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Week 40,n=2,0,0,0,0,6 | -0.5 (0.71) |  |  |  |  | 1.2 (0.75)

6. Primary Outcome: Change From Baseline in Mean Corpuscle Hemoglobin (MCH)
Description: Blood samples were collected at indicated time-points for analysis of hematology parameters like MCH. Baseline was defined as latest pre-dose assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 2, 3, 4 and 5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32, 36 and 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Picograms
  Day 2,n=12,6,6,9,9,6 | 0.03 (0.588) | 0.23 (0.388) | 0.02 (0.299) | -0.04 (0.255) | -0.02 (0.277) | -0.07 (0.450)
  Day 3,n=12,6,6,9,9,6 | 0.13 (0.485) | 0.25 (0.389) | 0.10 (0.283) | -0.02 (0.228) | 0.20 (0.444) | -0.08 (0.172)
  Day 4,n=12,6,6,8,8,6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 8 | 6
  Day 4,n=12,6,6,8,8,6 | 0.14 (0.542) | 0.17 (0.480) | 0.18 (0.299) | 0.05 (0.351) | 0.01 (0.432) | 0.12 (0.325)
  Day 5,n=12,6,6,9,9,6 | 0.08 (0.626) | 0.17 (0.314) | 0.22 (0.449) | -0.03 (0.346) | 0.02 (0.331) | -0.22 (0.240)
  Week 1,n=12,6,6,9,9,5: number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 5
  Week 1,n=12,6,6,9,9,5 | -0.07 (0.433) | 0.38 (0.542) | -0.07 (0.273) | 0.00 (0.381) | 0.00 (0.427) | -0.08 (0.553)
  Week 2,n=12,6,6,9,9,6 | -0.02 (0.495) | 0.33 (0.516) | 0.25 (0.418) | -0.08 (0.331) | -0.04 (0.088) | -0.02 (0.240)
  Week 4,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Week 4,n=12,6,5,9,9,6 | 0.15 (1.153) | 0.30 (0.374) | 0.12 (0.268) | -0.29 (0.404) | -0.06 (0.394) | -0.22 (0.343)
  Week 8,n=12,6,6,9,9,6 | -0.06 (0.429) | 0.25 (0.860) | 0.30 (0.410) | -0.30 (0.287) | -0.11 (0.655) | -0.22 (0.286)
  Week 12,n=12,6,6,9,9,5: number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 5
  Week 12,n=12,6,6,9,9,5 | -0.08 (0.583) | 0.32 (0.882) | 0.02 (0.624) | -0.42 (0.415) | -0.04 (0.541) | -0.60 (0.561)
  Week 18,n=12,6,6,9,9,6 | -0.13 (0.805) | 0.78 (0.382) | -0.10 (0.616) | -0.37 (0.384) | 0.01 (0.627) | -0.78 (0.382)
  Week 24,n=11,6,6,9,9,6: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 6
  Week 24,n=11,6,6,9,9,6 | -0.44 (0.883) | 0.87 (0.799) | 0.23 (0.356) | -0.37 (0.510) | -0.37 (0.632) | -0.90 (0.237)
  Week 26,n=12,6,6,9,9,6 | -0.27 (0.946) | 1.05 (0.505) | 0.10 (0.473) | -0.38 (0.432) | -0.71 (0.818) | -1.07 (0.393)
  Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Week 32,n=6,6,6,0,0,6 | 0.22 (0.975) | 0.67 (0.625) | 0.53 (0.909) |  |  | -0.58 (0.331)
  Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Week 36,n=6,0,0,9,9,0 | -1.00 (0.525) |  |  | -1.00 (0.403) | -0.68 (0.438) |
  Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Week 40,n=2,0,0,0,0,6 | -0.55 (0.071) |  |  |  |  | -0.68 (0.232)

7. Primary Outcome: Change From Baseline in Hemoglobin
Description: Blood samples were collected at indicated time-points for analysis of hematology parameters like hemoglobin. Baseline was defined as latest pre-dose assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 2, 3, 4 and 5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32, 36 and 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Grams per liter
  Day 2,n=12,6,6,9,9,6 | -2.4 (6.83) | 0.3 (6.80) | 3.7 (7.09) | -0.4 (6.00) | 4.3 (7.12) | 0.2 (8.52)
  Day 3,n=12,6,6,9,9,6 | 1.6 (6.78) | -0.5 (4.04) | 5.8 (8.80) | 0.1 (6.62) | 2.2 (4.35) | -0.5 (5.82)
  Day 4,n=12,6,6,8,8,6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 8 | 6
  Day 4,n=12,6,6,8,8,6 | -0.8 (6.69) | -1.3 (4.59) | 3.7 (6.02) | -1.0 (4.14) | 1.4 (5.32) | 3.2 (5.12)
  Day 5,n=12,6,6,9,9,6 | -5.0 (4.65) | -4.8 (3.82) | -0.3 (7.84) | -2.9 (4.54) | 0.8 (8.86) | -0.3 (5.13)
  Week 1,n=12,6,6,9,9,6 | -4.9 (6.50) | -8.3 (5.28) | 0.2 (6.79) | -1.4 (7.00) | 2.0 (6.42) | -1.5 (3.27)
  Week 2,n=12,6,6,9,9,6 | -3.3 (5.79) | -6.2 (4.67) | -3.7 (5.72) | -2.4 (6.29) | 3.3 (7.73) | -3.5 (6.50)
  Week 4,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Week 4,n=12,6,5,9,9,6 | -4.2 (5.08) | -8.0 (4.10) | -3.0 (7.94) | -4.2 (6.61) | 2.6 (10.36) | -2.5 (4.09)
  Week 8,n=12,6,6,9,9,6 | -1.1 (8.83) | -4.8 (4.96) | 1.5 (8.71) | -5.6 (6.27) | 4.9 (7.80) | -0.2 (2.48)
  Week 12,n=12,6,6,9,9,5: number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 5
  Week 12,n=12,6,6,9,9,5 | -4.3 (6.50) | -4.8 (4.49) | -0.2 (9.28) | -2.8 (7.98) | 5.9 (6.39) | -3.6 (2.07)
  Week 18,n=12,6,6,9,9,6 | -1.6 (8.47) | -1.8 (6.77) | -2.3 (6.62) | -2.4 (6.09) | 8.3 (9.25) | 0.5 (4.72)
  Week 24,n=11,6,6,9,9,6: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 6
  Week 24,n=11,6,6,9,9,6 | -5.3 (8.31) | -3.2 (7.99) | 0.5 (6.09) | -1.7 (6.36) | 2.4 (7.67) | -0.2 (3.37)
  Week 26,n=12,6,6,9,9,6 | -4.6 (9.70) | -4.5 (8.07) | -1.0 (5.76) | -2.2 (3.42) | 2.9 (6.23) | -2.7 (4.32)
  Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Week 32,n=6,6,6,0,0,6 | -1.7 (3.78) | -1.8 (4.79) | 5.2 (8.38) |  |  | -1.8 (5.71)
  Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Week 36,n=6,0,0,9,9,0 | -1.8 (8.47) |  |  | -2.4 (3.13) | 6.9 (10.67) |
  Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Week 40,n=2,0,0,0,0,6 | -3.5 (3.54) |  |  |  |  | -0.2 (4.17)

8. Primary Outcome: Change From Baseline in Hematocrit
Description: Blood samples were collected at indicated time-points for analysis of hematology parameters like hematocrit. Baseline was defined as latest pre-dose assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 2, 3, 4 and 5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32, 36 and 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Proportion of red blood cells in blood
  Day 2,n=12,6,6,9,9,6 | -0.007 (0.01961) | -0.001 (0.01884) | 0.009 (0.02262) | 0.000 (0.01500) | 0.011 (0.02356) | 0.007 (0.02689)
  Day 3,n=12,6,6,9,9,6 | 0.005 (0.01925) | -0.007 (0.01374) | 0.014 (0.02667) | 0.001 (0.01634) | -0.000 (0.01198) | 0.001 (0.01584)
  Day 4,n=12,6,6,8,8,6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 8 | 6
  Day 4,n=12,6,6,8,8,6 | -0.003 (0.01777) | -0.009 (0.01803) | 0.005 (0.02170) | -0.003 (0.01663) | -0.004 (0.01858) | 0.008 (0.01251)
  Day 5,n=12,6,6,9,9,6 | -0.010 (0.01509) | -0.015 (0.01340) | -0.004 (0.02743) | 0.001 (0.01970) | -0.001 (0.03295) | 0.006 (0.01061)
  Week 1,n=12,6,6,9,9,6 | -0.014 (0.01894) | -0.034 (0.01549) | 0.000 (0.02138) | -0.008 (0.02644) | -0.001 (0.02068) | -0.005 (0.01076)
  Week 2,n=12,6,6,9,9,6 | -0.010 (0.01670) | -0.025 (0.01626) | -0.016 (0.01928) | -0.009 (0.01960) | 0.002 (0.02469) | -0.011 (0.01759)
  Week 4,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Week 4,n=12,6,5,9,9,6 | -0.011 (0.01840) | -0.032 (0.01393) | -0.010 (0.02192) | -0.010 (0.02063) | 0.001 (0.02962) | -0.004 (0.01315)
  Week 8,n=12,6,6,9,9,6 | -0.001 (0.02285) | -0.020 (0.02119) | -0.000 (0.02367) | -0.011 (0.01889) | 0.005 (0.03084) | 0.002 (0.00750)
  Week 12,n=12,6,6,9,9,5: number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 5
  Week 12,n=12,6,6,9,9,5 | -0.010 (0.01745) | -0.025 (0.01262) | -0.001 (0.02587) | -0.005 (0.02379) | 0.006 (0.02343) | -0.006 (0.01279)
  Week 18,n=12,6,6,9,9,6 | -0.004 (0.02680) | -0.020 (0.02140) | -0.005 (0.03041) | -0.010 (0.02016) | 0.012 (0.02972) | 0.008 (0.01515)
  Week 24,n=11,6,6,9,9,6: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 6
  Week 24,n=11,6,6,9,9,6 | -0.013 (0.02108) | -0.023 (0.02325) | 0.001 (0.01955) | -0.006 (0.01726) | 0.001 (0.02607) | 0.009 (0.01184)
  Week 26,n=12,6,6,9,9,6 | -0.013 (0.02378) | -0.029 (0.02593) | -0.004 (0.01813) | -0.007 (0.01424) | 0.008 (0.01829) | 0.006 (0.01091)
  Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Week 32,n=6,6,6,0,0,6 | -0.005 (0.01904) | -0.015 (0.02220) | 0.009 (0.02413) |  |  | 0.002 (0.01851)
  Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Week 36,n=6,0,0,9,9,0 | 0.001 (0.01862) |  |  | -0.001 (0.01237) | 0.022 (0.03464) |
  Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Week 40,n=2,0,0,0,0,6 | -0.004 (0.00495) |  |  |  |  | 0.016 (0.00816)

9. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter: High Sensitivity C-reactive Protein (hsCRP)
Description: Blood samples were collected at indicated time-points for analysis of clinical parameters like hsCRP. Baseline was defined as latest pre-dose assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 2, 3, 4 and 5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32, 36 and 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Milligrams per liter
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Milligrams per liter
  Day 2,n=12,6,6,9,9,6 | -0.3443 (0.44689) | -0.1217 (0.28604) | -0.7367 (0.90943) | -0.3178 (0.45880) | -1.0956 (1.50219) | -0.4867 (0.50816)
  Day 3,n=11,6,6,9,9,6: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 6
  Day 3,n=11,6,6,9,9,6 | -0.4376 (0.43692) | -0.1417 (0.25818) | -0.8200 (1.10247) | -0.4367 (0.71042) | -1.4100 (2.19445) | -0.4817 (0.53663)
  Day 4,n=12,6,6,9,9,6 | -0.4570 (0.42874) | -0.1917 (0.23095) | -0.8683 (1.21224) | -0.5356 (0.91155) | -1.5311 (2.32545) | -0.5867 (0.66476)
  Day 5,n=12,6,6,9,9,6 | -0.3953 (0.37761) | -0.0117 (0.31244) | -0.7150 (1.23395) | -0.5322 (0.95860) | -1.4289 (2.35532) | -0.5867 (0.77590)
  Week 1,n=11,6,6,9,9,6: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 6
  Week 1,n=11,6,6,9,9,6 | -0.2176 (0.37960) | 0.2183 (0.23086) | -0.3033 (1.32284) | -0.5772 (0.86704) | -1.3156 (2.57735) | -0.5717 (0.69534)
  Week 2,n=12,6,6,9,9,6 | 0.0638 (0.44620) | 0.0167 (0.21435) | -0.6967 (1.30606) | 0.1733 (0.86781) | 0.2478 (2.91047) | -0.0967 (0.50091)
  Week 4,n=12,6,6,9,9,6 | -0.1253 (0.55902) | 0.1433 (0.66069) | -0.6433 (1.28969) | -0.2689 (0.86847) | 2.6422 (11.57024) | -0.4317 (0.54653)
  Week 8,n=12,6,6,9,9,6 | 0.5955 (1.62268) | 1.2817 (1.79930) | -0.3633 (1.66310) | -0.0878 (0.61243) | -1.1656 (2.91829) | -0.2517 (0.74440)
  Week 12,n=12,6,6,9,9,6 | 0.1455 (1.29507) | -0.1033 (0.36784) | 0.1250 (0.61656) | 0.9089 (1.31831) | -0.4067 (3.85725) | 0.1000 (0.55274)
  Week 18,n=12,6,6,9,9,6 | 0.1538 (0.54412) | 0.1883 (0.22851) | 0.1317 (1.77035) | 0.0700 (1.19067) | -1.1267 (2.89881) | -0.3300 (0.53457)
  Week 24,n=12,6,6,9,9,6 | 0.1163 (1.06052) | 0.4383 (1.46248) | -0.6383 (1.36902) | 0.1356 (0.80296) | -0.7989 (3.36420) | -0.2142 (1.09332)
  Week 26,n=12,6,6,9,9,6 | 0.2438 (0.75525) | 1.6333 (3.95614) | -0.6383 (1.13732) | 0.3344 (0.53761) | -0.6933 (3.25344) | 0.2400 (0.76467)
  Week 32,n=6,5,6,0,0,6: number analyzed (Participants) | 6 | 5 | 6 | 0 | 0 | 6
  Week 32,n=6,5,6,0,0,6 | 0.6393 (1.03514) | 0.2860 (0.82509) | -0.2400 (1.63862) |  |  | -0.1367 (0.73277)
  Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Week 36,n=6,0,0,9,9,0 | 0.4917 (1.31750) |  |  | -0.5456 (1.15831) | -0.1911 (3.93159) |
  Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Week 40,n=2,0,0,0,0,6 | -0.1450 (0.00707) |  |  |  |  | 0.4333 (1.74105)

10. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter of Total Protein and Albumin
Description: Blood samples were collected at indicated time-points for analysis of clinical parameters like total protein and albumin. Baseline was defined as latest pre-dose assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 2, 3, 4 and 5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32, 36 and 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Grams per liter
  Total protein, Day 2,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Total protein, Day 2,n=12,6,5,9,9,6 | -2.8 (3.74) | -2.3 (1.97) | -0.6 (3.36) | -3.8 (3.56) | 0.7 (4.90) | -0.2 (4.40)
  Total protein, Day 3,n=12,6,6,9,9,6 | -1.4 (3.68) | -2.5 (2.17) | 0.2 (3.43) | -1.7 (4.18) | -0.7 (3.16) | 0.0 (3.22)
  Total protein, Day 4,n=12,6,6,9,9,6 | -1.8 (4.34) | -1.2 (2.14) | 0.3 (2.58) | -2.8 (3.46) | -0.4 (2.65) | 1.7 (2.88)
  Total protein, Day 5,n=12,6,6,9,9,6 | -3.3 (2.77) | -2.7 (2.58) | -0.7 (4.72) | -3.2 (4.02) | 0.1 (5.78) | 0.0 (3.41)
  Total protein, Week 1,n=11,6,6,9,9,5: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 5
  Total protein, Week 1,n=11,6,6,9,9,5 | -1.6 (2.87) | -2.3 (4.23) | -2.8 (2.99) | -1.2 (4.29) | -1.1 (3.62) | -1.4 (1.95)
  Total protein, Week 2,n=12,6,6,9,9,6 | -1.8 (3.28) | -2.8 (4.26) | -2.8 (2.99) | -1.2 (4.29) | 1.1 (4.08) | -1.0 (3.58)
  Total protein, Week 4,n=12,6,6,9,9,6 | -2.5 (3.48) | -3.3 (3.01) | -0.8 (5.19) | -1.4 (3.09) | -0.1 (4.78) | -1.0 (3.41)
  Total protein, Week 8,n=12,6,6,9,9,6 | -1.0 (4.33) | -0.8 (5.15) | 0.2 (4.54) | -3.0 (3.94) | 1.4 (3.75) | 1.2 (3.37)
  Total protein, Week 12,n=12,6,6,9,9,6 | -2.8 (2.67) | -3.5 (4.59) | -0.5 (3.62) | -2.6 (3.71) | 2.7 (2.78) | 0.0 (2.10)
  Total protein, Week 18,n=12,6,6,9,9,6 | -1.3 (2.56) | -1.8 (5.23) | -1.7 (3.20) | -2.0 (3.64) | 1.7 (3.50) | 1.5 (3.08)
  Total protein, Week 24,n=12,6,6,9,9,6 | -3.3 (3.79) | -2.8 (4.54) | -1.0 (3.35) | -2.7 (3.04) | 0.6 (3.71) | 0.3 (2.73)
  Total protein, Week 26,n=12,6,6,9,9,6 | -2.5 (3.55) | -3.5 (2.88) | -2.3 (3.39) | -3.7 (1.87) | 1.0 (2.40) | 0.3 (2.34)
  Total protein, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Total protein, Week 32,n=6,6,6,0,0,6 | -1.7 (3.93) | 0.0 (3.63) | 0.3 (5.09) |  |  | -0.7 (2.66)
  Total protein, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Total protein, Week 36,n=6,0,0,9,9,0 | -1.5 (4.51) |  |  | -2.6 (3.21) | 1.8 (3.77) |
  Total protein, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Total protein, Week 40,n=2,0,0,0,0,6 | -2.5 (3.54) |  |  |  |  | 0.7 (1.63)
  Albumin, Day 2,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Albumin, Day 2,n=12,6,5,9,9,6 | -2.1 (2.68) | -1.3 (2.42) | -1.6 (2.07) | -2.4 (2.01) | -0.6 (3.36) | -0.5 (3.39)
  Albumin, Day 3,n=12,6,6,9,9,6 | -0.8 (2.70) | -1.3 (1.97) | -0.2 (2.48) | -1.4 (2.83) | -1.3 (2.06) | -0.3 (2.07)
  Albumin, Day 4,n=12,6,6,9,9,6 | -1.3 (2.63) | -0.5 (1.22) | -0.7 (1.86) | -2.2 (2.33) | -1.4 (1.81) | 0.3 (2.16)
  Albumin, Day 5,n=12,6,6,9,9,6 | -1.6 (1.68) | -1.5 (1.87) | -0.8 (3.54) | -2.3 (2.50) | -0.2 (3.49) | -0.2 (2.56)
  Albumin, Week 1,n=11,6,6,9,9,5: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 5
  Albumin, Week 1,n=11,6,6,9,9,5 | -0.5 (2.34) | -0.2 (2.86) | 0.0 (2.68) | -2.2 (2.28) | -1.4 (2.07) | -1.4 (2.97)
  Albumin, Week 2,n=12,6,6,9,9,6 | -0.8 (2.25) | -0.2 (1.83) | -1.7 (2.16) | -0.8 (2.86) | 0.4 (1.88) | -0.5 (1.52)
  Albumin, Week 4,n=12,6,6,9,9,6 | -1.8 (2.42) | -1.0 (2.28) | -0.3 (2.88) | -1.3 (1.87) | -0.6 (2.19) | -1.3 (2.73)
  Albumin, Week 8,n=12,6,6,9,9,6 | -0.8 (2.73) | -0.3 (2.88) | 0.7 (2.94) | -2.0 (2.69) | 0.7 (2.83) | 0.7 (2.34)
  Albumin, Week 12,n=12,6,6,9,9,6 | -1.5 (1.73) | -1.3 (2.80) | 0.0 (2.45) | -1.7 (2.40) | 0.4 (1.33) | -0.2 (2.32)
  Albumin, Week 18,n=12,6,6,9,9,6 | -0.5 (2.35) | -0.3 (2.94) | -1.5 (1.64) | -0.7 (2.06) | 0.2 (2.44) | 0.2 (1.94)
  Albumin, Week 24,n=12,6,6,9,9,6 | -1.7 (2.19) | 0.3 (2.73) | -0.8 (2.32) | -2.0 (1.87) | 0.4 (2.79) | -0.2 (2.04)
  Albumin, Week 26,n=12,6,6,9,9,6 | -1.6 (2.27) | -0.8 (1.72) | -1.8 (2.93) | -2.1 (0.60) | 0.1 (1.69) | -0.3 (2.07)
  Albumin, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Albumin, Week 32,n=6,6,6,0,0,6 | -0.5 (3.02) | 1.2 (3.06) | -0.2 (2.93) |  |  | -0.8 (2.14)
  Albumin, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Albumin, Week 36,n=6,0,0,9,9,0 | -0.7 (2.94) |  |  | -1.4 (1.67) | 0.6 (2.40) |
  Albumin, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Albumin, Week 40,n=2,0,0,0,0,6 | -1.0 (2.83) |  |  |  |  | -0.3 (1.63)

11. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters Like Total Bilirubin, Direct Bilirubin and Creatinine
Description: Blood samples were collected at indicated time-points for analysis of clinical parameters like total bilirubin, direct bilirubin and creatinine. Baseline was defined as latest pre-dose assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 2, 3, 4 and 5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32, 36 and 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Micromoles per liter
  Total bilirubin, Day 2,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Total bilirubin, Day 2,n=12,6,5,9,9,6 | -0.8 (3.86) | -1.3 (3.27) | -1.6 (4.34) | -0.2 (3.23) | 0.0 (5.20) | 1.0 (3.03)
  Total bilirubin, Day 3,n=12,6,6,9,9,6 | -1.3 (3.45) | -1.7 (3.44) | -1.7 (4.97) | 0.2 (3.80) | -0.4 (4.77) | 0.3 (2.34)
  Total bilirubin, Day 4,n=12,6,6,9,9,6 | -1.0 (3.13) | -2.7 (5.01) | -2.0 (7.48) | 0.0 (4.47) | 0.0 (4.47) | 1.0 (3.29)
  Total bilirubin, Day 5,n=12,6,6,9,9,6 | -2.3 (4.58) | -5.0 (5.76) | -2.0 (3.58) | -0.9 (5.49) | -1.3 (2.45) | -0.7 (3.27)
  Total bilirubin, Week 1,n=11,6,6,9,9,5: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 5
  Total bilirubin, Week 1,n=11,6,6,9,9,5 | -1.5 (4.82) | -0.7 (4.50) | 1.7 (1.97) | -1.1 (4.91) | 0.4 (3.84) | -2.0 (2.83)
  Total bilirubin, Week 2,n=12,6,6,9,9,6 | -1.2 (3.46) | -2.3 (6.12) | 0.7 (2.73) | 2.2 (2.91) | 0.4 (5.55) | 0.7 (2.42)
  Total bilirubin, Week 4,n=12,6,6,9,9,6 | -0.7 (2.15) | 0.3 (2.34) | 0.3 (1.97) | 0.0 (2.45) | -0.4 (5.81) | 1.0 (2.76)
  Total bilirubin, Week 8,n=12,6,6,9,9,6 | -1.2 (4.04) | -1.0 (6.29) | 2.0 (2.83) | 2.2 (4.06) | 0.4 (5.46) | -1.0 (4.69)
  Total bilirubin, Week 12,n=12,6,6,9,9,6 | -1.3 (4.03) | 0.0 (2.19) | 4.3 (5.85) | -0.9 (2.03) | 0.0 (4.69) | -0.7 (4.50)
  Total bilirubin, Week 18,n=12,6,6,9,9,6 | -0.3 (3.70) | -1.3 (6.53) | 2.0 (2.83) | 0.7 (1.73) | 0.4 (6.23) | -1.0 (3.52)
  Total bilirubin, Week 24,n=12,6,6,9,9,6 | -0.8 (4.47) | -1.3 (3.27) | 1.7 (3.88) | 0.2 (2.54) | 1.6 (6.98) | 2.0 (4.56)
  Total bilirubin, Week 26,n=12,6,6,9,9,6 | -1.3 (4.70) | 2.7 (3.93) | 0.3 (3.88) | -0.2 (3.80) | -0.7 (4.12) | 1.7 (2.34)
  Total bilirubin, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Total bilirubin, Week 32,n=6,6,6,0,0,6 | 0.7 (2.07) | -1.0 (5.62) | 0.0 (5.22) |  |  | 0.0 (4.90)
  Total bilirubin, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Total bilirubin, Week 36,n=6,0,0,9,9,0 | -0.7 (7.12) |  |  | 0.4 (3.13) | -1.1 (5.67) |
  Total bilirubin, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Total bilirubin, Week 40,n=2,0,0,0,0,6 | 2.0 (0.00) |  |  |  |  | 0.7 (2.07)
  Direct bilirubin, Day 2,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Direct bilirubin, Day 2,n=12,6,5,9,9,6 | -0.3 (1.15) | -0.7 (1.03) | -0.4 (0.89) | -0.2 (1.20) | 0.2 (1.20) | 0.3 (0.82)
  Direct bilirubin, Day 3,n=12,6,6,9,9,6 | -0.5 (0.90) | -0.3 (0.82) | -0.3 (0.82) | 0.4 (1.67) | 0.0 (1.00) | 0.0 (1.26)
  Direct bilirubin, Day 4,n=12,6,6,9,9,6 | -0.5 (0.90) | -0.3 (0.82) | -0.7 (1.03) | 0.2 (1.56) | 0.2 (1.20) | -0.3 (0.82)
  Direct bilirubin, Day 5,n=12,6,6,9,9,6 | -0.7 (0.98) | -0.7 (1.03) | -0.7 (1.03) | 0.2 (1.56) | 0.0 (1.00) | -0.7 (1.03)
  Direct bilirubin, Week 1,n=11,6,6,9,9,5: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 5
  Direct bilirubin, Week 1,n=11,6,6,9,9,5 | -0.5 (0.93) | -0.3 (0.82) | -0.3 (0.82) | 0.0 (1.41) | 0.0 (1.00) | -0.8 (1.10)
  Direct bilirubin, Week 2,n=12,6,6,9,9,6 | -0.3 (1.15) | 0.0 (0.00) | 0.0 (0.00) | 0.7 (1.41) | 0.2 (1.20) | 0.3 (1.51)
  Direct bilirubin, Week 4,n=12,6,6,9,9,6 | 0.0 (0.85) | 0.0 (1.26) | 0.3 (0.82) | 0.2 (1.20) | 0.2 (1.20) | 0.0 (1.26)
  Direct bilirubin, Week 8,n=12,6,6,9,9,6 | -0.2 (1.03) | 0.0 (0.00) | 0.3 (0.82) | 0.9 (1.45) | 0.4 (1.33) | -0.7 (1.03)
  Direct bilirubin, Week 12,n=12,6,6,9,9,6 | -0.5 (0.90) | 0.0 (1.26) | 0.3 (0.82) | 0.2 (1.20) | 0.2 (1.20) | -0.3 (1.51)
  Direct bilirubin, Week 18,n=12,6,6,9,9,6 | -0.2 (1.03) | 0.0 (1.26) | 0.0 (0.00) | 0.7 (1.00) | 0.4 (1.33) | 0.0 (1.26)
  Direct bilirubin, Week 24,n=12,6,6,9,9,6 | -0.3 (0.78) | 0.3 (1.51) | -0.3 (0.82) | 0.2 (1.20) | 0.9 (1.76) | 0.0 (1.26)
  Direct bilirubin, Week 26,n=12,6,6,9,9,6 | 0.0 (1.21) | 0.7 (1.03) | 0.3 (0.82) | 0.0 (1.41) | 0.0 (1.00) | 0.0 (1.26)
  Direct bilirubin, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Direct bilirubin, Week 32,n=6,6,6,0,0,6 | -0.3 (0.82) | -0.3 (0.82) | -0.3 (1.51) |  |  | 0.0 (1.26)
  Direct bilirubin, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Direct bilirubin, Week 36,n=6,0,0,9,9,0 | 0.0 (1.79) |  |  | 0.0 (1.00) | 0.4 (1.67) |
  Direct bilirubin, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Direct bilirubin, Week 40,n=2,0,0,0,0,6 | -1.0 (1.41) |  |  |  |  | -0.3 (0.82)
  Creatinine, Day 2,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Creatinine, Day 2,n=12,6,5,9,9,6 | -2.80 (5.501) | -1.03 (3.930) | -1.42 (3.512) | -4.91 (4.835) | -0.77 (4.863) | -1.63 (6.417)
  Creatinine, Day 3,n=12,6,6,9,9,6 | -3.48 (6.036) | -1.78 (3.571) | -2.95 (6.208) | -1.58 (4.913) | -1.87 (5.026) | -1.20 (3.795)
  Creatinine, Day 4,n=12,6,6,9,9,6 | 0.29 (6.544) | -0.73 (4.126) | -0.75 (7.123) | -4.64 (6.296) | -0.88 (3.180) | 3.68 (7.962)
  Creatinine, Day 5,n=12,6,6,9,9,6 | -2.73 (5.166) | 0.72 (1.883) | -2.53 (4.541) | -4.63 (6.355) | 0.39 (3.085) | -1.62 (5.216)
  Creatinine, Week 1,n=11,6,6,9,9,5: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 5
  Creatinine, Week 1,n=11,6,6,9,9,5 | -2.49 (7.084) | 3.68 (4.892) | -2.08 (6.098) | -3.06 (6.393) | 0.59 (4.303) | -0.70 (7.736)
  Creatinine, Week 2,n=12,6,6,9,9,6 | -1.12 (5.854) | 1.47 (5.019) | -0.90 (6.377) | -2.67 (5.702) | 2.27 (5.322) | 0.73 (7.868)
  Creatinine, Week 4,n=12,6,6,9,9,6 | -1.28 (4.730) | -2.80 (3.839) | 0.27 (3.837) | 0.09 (6.843) | 0.59 (5.989) | 6.05 (6.066)
  Creatinine, Week 8,n=12,6,6,9,9,6 | -1.40 (6.462) | 0.28 (5.062) | -1.20 (7.277) | 0.19 (3.718) | 6.00 (4.511) | 1.63 (4.317)
  Creatinine, Week 12,n=12,6,6,9,9,6 | -0.30 (7.643) | 0.88 (5.043) | 1.03 (5.846) | -0.41 (4.748) | 5.01 (3.820) | 0.72 (4.532)
  Creatinine, Week 18,n=12,6,6,9,9,6 | -1.27 (7.753) | 1.75 (4.831) | 2.05 (7.131) | 2.83 (5.033) | 4.42 (5.191) | 1.15 (6.297)
  Creatinine, Week 24,n=12,6,6,9,9,6 | 0.89 (4.393) | 1.77 (5.597) | 1.60 (5.877) | 7.07 (6.581) | 2.66 (6.005) | 2.20 (4.431)
  Creatinine, Week 26,n=12,6,6,9,9,6 | -2.29 (5.633) | -2.22 (5.017) | 0.27 (15.342) | 3.16 (6.620) | 0.69 (3.857) | 3.22 (5.653)
  Creatinine, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Creatinine, Week 32,n=6,6,6,0,0,6 | 0.00 (5.871) | 0.87 (5.904) | 6.60 (6.880) |  |  | 2.05 (2.474)
  Creatinine, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Creatinine, Week 36,n=6,0,0,9,9,0 | -0.60 (4.767) |  |  | 2.57 (4.347) | 10.42 (6.864) |
  Creatinine, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Creatinine, Week 40,n=2,0,0,0,0,6 | 1.75 (2.475) |  |  |  |  | 1.60 (6.174)

12. Primary Outcome: Urine Specific Gravity Analysis by Dipstick Method
Description: Urinary specific gravity measurement is a routine part of urinalysis. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity.
Time Frame: Baseline and at Days 2, 3, 4 and 5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32, 36 and 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 1
Ratio
  Day 2,n=1,2,0,2,0,0: number analyzed (Participants) | 1 | 2 | 0 | 2 | 0 | 0
  Day 2,n=1,2,0,2,0,0 | 1.0200 (NA) — NA indicates that standard deviation could not be calculated for a single data point. | 1.0125 (0.00354) |  | 1.0120 (0.00283) |  |
  Day 3,n=2,0,0,1,0,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0 | 0
  Day 3,n=2,0,0,1,0,0 | 1.0265 (0.00212) |  |  | 1.0280 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |  |
  Day 4,n=0,0,1,1,0,0: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 0
  Day 4,n=0,0,1,1,0,0 |  |  | 1.0150 (NA) — NA indicates that standard deviation could not be calculated for a single data point. | 1.0290 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |  |
  Day 5,n=2,0,0,2,1,0: number analyzed (Participants) | 2 | 0 | 0 | 2 | 1 | 0
  Day 5,n=2,0,0,2,1,0 | 1.0275 (0.00354) |  |  | 1.0205 (0.00919) | 1.0140 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |
  Week 1,n=2,1,1,3,0,0: number analyzed (Participants) | 2 | 1 | 1 | 3 | 0 | 0
  Week 1,n=2,1,1,3,0,0 | 1.0235 (0.00212) | 1.0260 (NA) — NA indicates that standard deviation could not be calculated for a single data point. | 1.0250 (NA) — NA indicates that standard deviation could not be calculated for a single data point. | 1.0197 (0.00751) |  |
  Week 2,n=1,0,0,4,1,0: number analyzed (Participants) | 1 | 0 | 0 | 4 | 1 | 0
  Week 2,n=1,0,0,4,1,0 | 1.0250 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |  |  | 1.0218 (0.00822) | 1.0130 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |
  Week 4,n=3,1,1,5,0,1: number analyzed (Participants) | 3 | 1 | 1 | 5 | 0 | 1
  Week 4,n=3,1,1,5,0,1 | 1.0193 (0.00839) | 1.0150 (NA) — NA indicates that standard deviation could not be calculated for a single data point. | 1.0250 (NA) — NA indicates that standard deviation could not be calculated for a single data point. | 1.0158 (0.01052) |  | 1.0270 (NA) — NA indicates that standard deviation could not be calculated for a single data point.
  Week 8,n=1,0,0,2,0,0: number analyzed (Participants) | 1 | 0 | 0 | 2 | 0 | 0
  Week 8,n=1,0,0,2,0,0 | 1.0300 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |  |  | 1.0220 (0.00566) |  |
  Week 12,n=0,1,0,1,0,0: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 0
  Week 12,n=0,1,0,1,0,0 |  | 1.0180 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |  | 1.0230 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |  |
  Week 18,n=3,1,0,1,0,0: number analyzed (Participants) | 3 | 1 | 0 | 1 | 0 | 0
  Week 18,n=3,1,0,1,0,0 | 1.0260 (0.00265) | 1.0180 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |  | 1.0230 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |  |
  Week 24,n=1,1,0,4,0,0: number analyzed (Participants) | 1 | 1 | 0 | 4 | 0 | 0
  Week 24,n=1,1,0,4,0,0 | 1.0200 (NA) — NA indicates that standard deviation could not be calculated for a single data point. | 1.0230 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |  | 1.0200 (0.00374) |  |
  Week 26,n=0,0,0,2,0,0: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0
  Week 26,n=0,0,0,2,0,0 |  |  |  | 1.0240 (0.00566) |  |
  Week 32,n=1,0,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Week 32,n=1,0,0,0,0,0 | 1.0150 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |  |  |  |  |
  Week 36,n=0,0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Week 40,n=0,0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were assessed in a supine position after 5 minutes of rest. Baseline was defined as latest pre-dose assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at 2 and 8 hours at Day 1; Days 2, 3, 4 and 5; Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32, 36 and 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Millimeters of mercury
  SBP, 2 hours Day1,n=12,6,6,9,9,6 | -0.3 (6.08) | -2.2 (7.47) | 3.3 (7.37) | -0.9 (7.18) | -1.8 (7.19) | -2.0 (8.58)
  SBP, 8 hours Day1,n=12,6,6,9,9,6 | 0.0 (6.00) | 4.2 (10.01) | 3.0 (8.46) | 1.7 (10.69) | 4.9 (7.52) | -2.2 (5.64)
  SBP, Day 2,n=12,6,6,9,9,6 | -2.5 (7.00) | -0.8 (8.08) | 6.0 (4.86) | 1.8 (9.11) | 6.3 (7.42) | -5.3 (4.37)
  SBP, Day 3,n=12,6,6,9,9,6 | 2.6 (9.21) | -2.2 (7.36) | 3.7 (9.16) | 1.0 (10.68) | -0.1 (4.43) | -5.0 (6.00)
  SBP, Day 4,n=12,6,6,9,9,6 | 0.8 (5.75) | -2.2 (6.24) | 2.3 (8.09) | 0.3 (6.91) | 2.9 (6.86) | -3.3 (7.39)
  SBP, Day 5,n=12,6,6,9,9,6 | -3.0 (6.05) | 0.8 (6.82) | 1.0 (7.72) | -2.8 (9.81) | 0.4 (3.91) | -4.7 (4.46)
  SBP, Week 1,n=12,6,6,9,9,6 | -0.3 (8.86) | 0.3 (7.50) | 1.5 (6.60) | -2.7 (9.06) | 1.7 (5.02) | 0.2 (8.13)
  SBP, Week 2,n=12,6,6,9,9,6 | -2.6 (5.90) | 1.0 (10.22) | 5.8 (5.85) | 4.2 (10.45) | 0.8 (11.04) | -2.8 (9.83)
  SBP, Week 4,n=12,6,6,9,9,6 | -1.6 (8.80) | 0.3 (8.82) | 7.0 (11.26) | 3.2 (14.09) | 0.9 (6.11) | -2.3 (7.15)
  SBP, Week 8,n=12,6,6,9,9,6 | 0.7 (9.71) | 0.0 (9.27) | 2.0 (12.66) | 3.1 (8.52) | -1.4 (6.60) | -1.8 (5.91)
  SBP, Week 12,n=12,6,6,9,9,6 | -0.8 (5.13) | 1.2 (5.19) | 2.3 (9.97) | 5.4 (9.41) | 0.0 (7.37) | -4.2 (11.18)
  SBP, Week 18,n=12,6,6,9,9,6 | -0.6 (6.86) | 4.2 (9.15) | 3.8 (13.33) | 2.0 (8.76) | 2.1 (9.52) | -7.3 (15.49)
  SBP, Week 24,n=12,6,6,9,9,6 | -0.8 (8.22) | 9.3 (10.42) | 3.7 (6.59) | 2.9 (9.91) | 1.9 (12.06) | -2.2 (6.46)
  SBP, Week 26,n=12,6,6,9,9,6 | 3.0 (11.95) | 3.2 (6.11) | 3.2 (5.91) | 7.9 (10.13) | 2.9 (7.56) | -5.8 (6.11)
  SBP, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  SBP, Week 32,n=6,6,6,0,0,6 | 3.0 (6.90) | -3.8 (12.45) | 8.7 (10.61) |  |  | -3.3 (6.89)
  SBP, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  SBP, Week 36,n=6,0,0,9,9,0 | -3.5 (13.72) |  |  | 2.8 (9.59) | 2.8 (7.77) |
  SBP, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  SBP, Week 40,n=2,0,0,0,0,6 | -15.0 (14.14) |  |  |  |  | -5.8 (17.52)
  DBP, 2 hours Day1,n=12,6,6,9,9,6 | -2.9 (5.00) | 3.3 (4.89) | 4.3 (9.14) | -2.2 (4.18) | -2.2 (6.14) | -3.8 (1.94)
  DBP, 8 hours Day1,n=12,6,6,9,9,6 | -0.6 (4.34) | 2.0 (7.46) | 0.5 (9.52) | -1.3 (4.58) | -2.0 (5.74) | -1.8 (5.56)
  DBP, Day 2,n=12,6,6,9,9,6 | -0.2 (4.47) | 0.8 (4.49) | 3.0 (5.83) | -1.1 (5.67) | 4.7 (4.18) | 0.0 (4.94)
  DBP, Day 3,n=12,6,6,9,9,6 | 0.6 (3.99) | -1.3 (7.26) | 3.0 (7.04) | -2.6 (5.41) | -0.3 (4.30) | -0.3 (6.44)
  DBP, Day 4,n=12,6,6,9,9,6 | -0.1 (5.04) | 2.3 (4.80) | -1.0 (5.69) | -0.2 (5.14) | 0.1 (3.76) | -2.8 (3.82)
  DBP, Day 5,n=12,6,6,9,9,6 | -1.4 (4.40) | 4.8 (6.49) | 0.7 (8.09) | -4.1 (7.29) | 0.9 (4.23) | -1.5 (2.81)
  DBP, Week 1,n=12,6,6,9,9,6 | 0.6 (5.37) | 3.7 (6.98) | 4.3 (9.27) | -0.4 (5.68) | 0.8 (3.38) | 0.0 (5.44)
  DBP, Week 2,n=12,6,6,9,9,6 | 1.1 (6.23) | 4.7 (5.65) | 6.0 (8.99) | 1.6 (4.36) | 1.9 (6.92) | 0.2 (4.62)
  DBP, Week 4,n=12,6,6,9,9,6 | 0.3 (6.17) | 1.3 (7.74) | 4.2 (11.36) | 3.1 (6.09) | 1.6 (5.41) | 3.8 (4.40)
  DBP, Week 8,n=12,6,6,9,9,6 | 1.3 (3.73) | 5.2 (5.49) | 5.5 (13.28) | 3.3 (4.95) | 0.7 (4.21) | 0.5 (3.94)
  DBP, Week 12,n=12,6,6,9,9,6 | 0.9 (6.29) | 3.2 (5.91) | 1.7 (14.15) | 3.4 (5.39) | 3.6 (4.72) | 1.3 (5.09)
  DBP, Week 18,n=12,6,6,9,9,6 | -2.1 (6.63) | 3.3 (5.68) | 3.0 (12.65) | 0.7 (6.84) | 3.8 (8.07) | 0.5 (7.50)
  DBP, Week 24,n=12,6,6,9,9,6 | -1.6 (7.77) | 6.3 (5.35) | 4.0 (9.78) | 5.3 (6.56) | 1.1 (9.12) | 2.0 (5.66)
  DBP, Week 26,n=12,6,6,9,9,6 | -0.5 (7.23) | 3.2 (4.36) | 3.8 (9.45) | 6.6 (8.38) | 1.8 (8.61) | 0.2 (3.97)
  DBP, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  DBP, Week 32,n=6,6,6,0,0,6 | 1.3 (2.34) | -0.2 (6.49) | 7.0 (4.34) |  |  | 2.0 (7.64)
  DBP, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  DBP, Week 36,n=6,0,0,9,9,0 | 2.3 (13.13) |  |  | 3.6 (5.64) | 2.3 (8.82) |
  DBP, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  DBP, Week 40,n=2,0,0,0,0,6 | 0.5 (4.95) |  |  |  |  | -3.5 (6.95)

14. Primary Outcome: Change From Baseline in Temperature
Description: Temperature was assessed in a supine position after 5 minutes of rest. Baseline was defined as latest pre-dose assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at 2 and 8 hours at Day 1; Days 2, 3, 4 and 5; Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32, 36 and 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Degree Celsius
  2 hours Day1,n=12,6,6,9,9,6 | 0.05 (0.419) | 0.32 (0.293) | 0.13 (0.163) | 0.30 (0.474) | 0.03 (0.328) | 0.00 (0.420)
  Category title 2. 8 hours Day1,n=12,6,6,9,9,6 | 0.13 (0.405) | 0.40 (0.410) | 0.07 (0.234) | 0.24 (0.513) | 0.18 (0.291) | 0.35 (0.589)
  Category title 3. Day 2,n=12,6,6,9,9,6 | -0.01 (0.312) | 0.23 (0.437) | 0.10 (0.429) | -0.03 (0.559) | -0.01 (0.333) | -0.05 (0.259)
  Day 3,n=12,6,6,9,9,6 | -0.10 (0.402) | 0.02 (0.538) | 0.02 (0.256) | 0.13 (0.439) | 0.02 (0.315) | 0.12 (0.343)
  Day 4,n=12,6,6,9,9,6 | -0.03 (0.260) | 0.15 (0.554) | 0.08 (0.293) | 0.11 (0.382) | 0.22 (0.239) | 0.02 (0.397)
  Day 5,n=12,6,6,9,9,6 | -0.08 (0.171) | 0.13 (0.516) | 0.25 (0.464) | -0.07 (0.300) | -0.04 (0.255) | 0.12 (0.293)
  Week 1,n=12,6,6,9,9,6 | -0.13 (0.293) | 0.32 (0.492) | 0.18 (0.147) | 0.12 (0.399) | 0.01 (0.359) | 0.18 (0.232)
  Week 2,n=12,6,6,9,9,6 | -0.29 (0.448) | 0.30 (0.460) | 0.03 (0.333) | 0.04 (0.340) | 0.08 (0.441) | -0.08 (0.319)
  Week 4,n=12,6,6,9,9,6 | -0.23 (0.172) | 0.20 (0.400) | -0.02 (0.387) | -0.09 (0.302) | 0.00 (0.671) | -0.03 (0.258)
  Week 8,n=12,6,6,9,9,6 | 0.00 (0.280) | 0.32 (0.397) | -0.18 (0.504) | 0.09 (0.446) | 0.02 (0.282) | 0.13 (0.197)
  Week 12,n=12,6,6,9,9,6 | -0.10 (0.386) | 0.17 (0.356) | -0.15 (0.187) | 0.09 (0.337) | -0.09 (0.355) | 0.00 (0.369)
  Week 18,n=12,6,6,9,9,6 | -0.07 (0.267) | 0.18 (0.662) | 0.02 (0.407) | 0.13 (0.512) | 0.07 (0.283) | -0.05 (0.399)
  Week 24,n=12,6,6,9,9,6 | -0.07 (0.396) | 0.08 (0.488) | 0.08 (0.319) | -0.02 (0.367) | -0.07 (0.316) | -0.02 (0.133)
  Week 26,n=12,6,6,9,9,6 | -0.08 (0.311) | 0.03 (0.441) | -0.02 (0.504) | 0.08 (0.424) | 0.00 (0.442) | -0.22 (0.117)
  Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Week 32,n=6,6,6,0,0,6 | -0.30 (0.569) | 0.48 (1.363) | 0.02 (0.306) |  |  | 0.08 (0.331)
  Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Week 36,n=6,0,0,9,9,0 | 0.22 (0.366) |  |  | 0.14 (0.433) | -0.03 (0.212) |
  Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Week 40,n=2,0,0,0,0,6 | -0.10 (0.566) |  |  |  |  | -0.05 (0.084)

15. Primary Outcome: Change From Baseline in Heart Rate
Description: Heart rate was assessed in a supine position after 5 minutes of rest. Baseline was defined as latest pre-dose assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at 2 and 8 hours at Day 1; Days 2, 3, 4 and 5; Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32, 36 and 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Beats per minute
  2 hours Day1,n=12,6,6,9,9,6 | 2.2 (13.62) | -4.2 (5.27) | -3.3 (8.64) | 0.8 (14.45) | 0.9 (10.74) | 5.2 (5.46)
  8 hours Day1,n=12,6,6,9,9,6 | -1.0 (7.05) | -2.0 (7.27) | -3.2 (3.37) | 0.3 (14.21) | 1.0 (11.62) | 4.8 (8.06)
  Day 2,n=12,6,6,9,9,6 | -1.2 (6.59) | -1.5 (2.81) | -1.7 (3.83) | -4.0 (11.03) | 2.7 (8.14) | -0.7 (3.50)
  Day 3,n=12,6,6,9,9,6 | -0.2 (4.82) | 0.2 (5.88) | 1.3 (8.41) | 0.7 (4.92) | 4.7 (3.94) | -1.0 (7.40)
  Day 4,n=12,6,6,9,9,6 | 3.8 (7.53) | 1.7 (4.84) | 4.7 (8.98) | -1.2 (11.62) | 3.6 (5.27) | 1.5 (3.33)
  Day 5,n=12,6,6,9,9,6 | 1.1 (4.91) | 2.8 (8.61) | 1.2 (7.83) | -0.1 (10.30) | 0.6 (4.28) | 3.0 (4.47)
  Week 1,n=12,6,6,9,9,6 | -1.8 (6.03) | 0.0 (10.58) | -1.8 (7.05) | -1.1 (10.80) | 1.4 (5.98) | 5.0 (9.21)
  Week 2,n=12,6,6,9,9,6 | -4.8 (5.57) | -1.3 (5.89) | -5.2 (5.23) | 2.1 (12.38) | 1.0 (10.51) | 2.0 (6.00)
  Week 4,n=12,6,6,9,9,6 | -3.2 (8.46) | -2.3 (2.88) | -1.5 (5.96) | -1.1 (10.54) | 0.8 (13.58) | 0.5 (9.35)
  Week 8,n=12,6,6,9,9,6 | -0.2 (7.12) | -1.8 (7.14) | -3.7 (5.79) | -4.9 (15.39) | -0.6 (6.52) | -0.3 (4.72)
  Week 12,n=12,6,6,9,9,6 | -1.2 (10.47) | 3.3 (8.38) | -2.3 (6.53) | 0.6 (16.41) | 1.0 (9.31) | 3.0 (7.38)
  Week 18,n=12,6,6,9,9,6 | -3.2 (8.56) | -2.0 (7.07) | -1.7 (5.50) | 0.8 (10.84) | 1.7 (9.10) | 2.5 (7.23)
  Week 24,n=12,6,6,9,9,6 | -1.4 (10.03) | -0.8 (6.85) | 1.8 (7.68) | -2.8 (12.04) | 3.2 (9.28) | 0.0 (4.82)
  Week 26,n=12,6,6,9,9,6 | -2.7 (10.04) | -0.2 (2.56) | -0.7 (6.59) | 2.0 (12.03) | 1.6 (7.09) | 1.8 (4.58)
  Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Week 32,n=6,6,6,0,0,6 | -1.0 (10.55) | -2.2 (5.19) | 0.7 (6.06) |  |  | 0.8 (7.28)
  Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Week 36,n=6,0,0,9,9,0 | 0.5 (11.59) |  |  | 0.0 (12.50) | 2.6 (6.29) |
  Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Week 40,n=2,0,0,0,0,6 | -2.0 (2.83) |  |  |  |  | 2.8 (10.26)

16. Primary Outcome: Change From Baseline in Respiration Rate
Description: Respiration rate was assessed in a supine position after 5 minutes of rest. Baseline was defined as latest pre-dose assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at 2 and 8 hours at Day 1; Days 2, 3, 4 and 5; Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32, 36 and 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Breaths per minute
  2 hours Day1,n=12,6,6,9,9,6 | 0.8 (2.42) | 1.2 (1.83) | 0.0 (2.53) | 0.3 (2.65) | 0.8 (1.72) | 2.2 (3.31)
  8 hours Day1,n=12,6,6,9,9,6 | -0.1 (2.19) | 0.5 (3.27) | -1.0 (1.79) | 1.0 (3.28) | 2.1 (1.83) | 0.3 (1.63)
  Day 2,n=12,6,6,9,9,6 | -0.7 (2.64) | 1.7 (2.58) | -1.2 (1.47) | 1.9 (1.96) | 1.8 (1.30) | 1.5 (2.07)
  Day 3,n=12,6,6,9,9,6 | -1.0 (2.83) | 1.5 (3.27) | -0.2 (2.40) | 1.1 (2.80) | 1.2 (2.11) | 0.7 (3.50)
  Day 4,n=12,6,6,9,9,6 | -0.1 (3.06) | -1.0 (3.03) | 0.7 (1.21) | 0.3 (2.24) | 2.3 (1.87) | 0.2 (2.71)
  Day 5,n=12,6,6,9,9,6 | -1.1 (2.39) | 0.7 (3.20) | -1.5 (1.05) | 0.0 (2.55) | 1.3 (2.18) | 0.0 (1.41)
  Week 1,n=12,6,6,9,9,6 | -0.5 (3.45) | 0.7 (3.67) | -0.2 (1.33) | -0.6 (1.67) | 0.4 (1.81) | -1.8 (2.71)
  Week 2,n=12,6,6,9,9,6 | -0.3 (2.15) | 0.7 (4.08) | 0.2 (2.23) | 1.1 (2.76) | 0.9 (2.98) | -0.2 (3.06)
  Week 4,n=12,6,6,9,9,6 | 0.5 (3.18) | 1.5 (2.59) | 1.5 (1.22) | 0.4 (1.88) | 1.2 (2.17) | -0.5 (3.89)
  Week 8,n=12,6,6,9,9,6 | -0.5 (2.71) | 0.5 (2.81) | 0.3 (2.42) | 0.1 (3.41) | 2.3 (2.18) | 0.7 (2.80)
  Week 12,n=12,6,6,9,9,6 | 0.0 (3.49) | 0.7 (4.63) | 0.7 (2.16) | 1.2 (2.86) | 0.9 (1.69) | -0.3 (2.88)
  Week 18,n=12,6,6,9,9,6 | 0.5 (3.66) | -0.2 (3.06) | -0.7 (1.97) | 1.4 (2.07) | 1.4 (1.42) | 1.2 (3.25)
  Week 24,n=12,6,6,9,9,6 | -0.8 (2.59) | -0.7 (4.41) | -0.7 (1.51) | 1.4 (2.13) | 0.7 (2.40) | 0.8 (1.94)
  Week 26,n=12,6,6,9,9,6 | -1.1 (2.43) | 0.5 (3.02) | -0.7 (1.51) | 0.6 (2.01) | 1.6 (2.19) | 0.3 (3.01)
  Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Week 32,n=6,6,6,0,0,6 | -1.5 (1.76) | 1.3 (3.01) | 0.7 (2.34) |  |  | 1.0 (3.10)
  Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Week 36,n=6,0,0,9,9,0 | 0.2 (1.83) |  |  | 0.2 (2.64) | 1.3 (1.50) |
  Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Week 40,n=2,0,0,0,0,6 | -2.0 (1.41) |  |  |  |  | -0.3 (1.86)

17. Primary Outcome: Change From Baseline in Heart Rate: Electrocardiogram (ECG)
Description: 12-lead ECG were performed in a supine position using an automated ECG machine that calculated the heart rate and measured PR, QRS, QT and corrected QT (QTc) intervals. ECG measurements were performed in triplicate. When multiple ECGs were performed at the same planned timepoint, the average value of each parameter was used. Baseline was defined as latest pre-dose assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at 2 and 8 hours on Day 1; Days 2, 3, 4 and 5; Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32, 36 and 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Beats per minute
  2 hours Day1,n=12,6,5,9,8,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 8 | 6
  2 hours Day1,n=12,6,5,9,8,6 | 1.4 (11.13) | -4.3 (7.81) | -4.6 (4.56) | 0.2 (11.06) | 0.3 (11.85) | 6.8 (7.01)
  8 hours Day1,n=12,6,6,9,9,6 | 0.1 (6.34) | -0.8 (8.93) | -6.3 (6.10) | -1.3 (6.23) | 0.0 (14.05) | 4.1 (6.20)
  Day 2,n=12,6,6,9,9,6 | 0.4 (4.68) | -0.4 (5.67) | 0.8 (5.29) | -1.4 (6.32) | -0.3 (7.34) | 0.3 (1.06)
  Day 3,n=12,6,6,9,9,6 | 1.5 (5.93) | 0.3 (4.15) | 0.4 (7.36) | 1.5 (7.03) | 3.1 (3.48) | 1.9 (3.69)
  Day 4,n=12,6,6,9,9,6 | 3.5 (5.11) | 1.5 (8.64) | 5.5 (9.13) | 3.1 (11.04) | 2.6 (4.60) | 3.2 (3.97)
  Day 5,n=12,6,6,9,9,6 | 1.8 (4.78) | 1.5 (9.63) | 0.8 (5.24) | 2.5 (5.29) | -0.4 (5.97) | 2.6 (4.75)
  Week 1,n=12,6,6,9,9,6 | -2.8 (5.74) | 1.6 (5.76) | -2.4 (5.53) | 2.4 (9.66) | 2.0 (4.76) | 4.9 (7.60)
  Week 2,n=12,6,6,9,9,6 | -4.2 (5.32) | -2.3 (5.02) | -5.9 (5.91) | 1.8 (10.26) | 1.7 (13.56) | 1.7 (7.11)
  Week 4,n=12,6,6,9,9,6 | -3.8 (7.01) | -1.6 (3.75) | -1.2 (3.45) | -1.6 (7.53) | -0.3 (14.55) | -0.9 (6.25)
  Week 8,n=12,6,6,9,9,6 | -0.8 (5.91) | -0.6 (6.22) | -2.0 (6.02) | -2.9 (7.50) | -0.7 (9.14) | 0.6 (4.97)
  Week 12,n=12,6,6,9,9,6 | 0.3 (11.83) | -1.3 (6.24) | -3.3 (6.35) | 1.8 (15.28) | 0.4 (11.55) | 1.3 (6.44)
  Week 18,n=12,6,6,9,9,6 | -3.4 (9.05) | -0.4 (6.59) | -3.3 (5.20) | 1.6 (6.92) | 0.6 (8.78) | 2.2 (4.65)
  Week 24,n=12,6,6,9,9,6 | -2.7 (7.95) | -0.2 (8.28) | 2.5 (8.00) | -0.3 (9.13) | 1.7 (11.03) | 1.2 (6.47)
  Week 26,n=12,6,6,9,9,6 | -2.0 (9.35) | -0.3 (5.16) | -1.5 (7.18) | 2.5 (11.97) | 2.0 (8.22) | 0.3 (7.66)
  Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Week 32,n=6,6,6,0,0,6 | -2.7 (9.21) | -4.6 (7.34) | 0.7 (5.84) |  |  | 2.3 (6.46)
  Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Week 36,n=6,0,0,9,9,0 | 1.5 (7.13) |  |  | -0.2 (10.26) | 1.3 (5.74) |
  Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Week 40,n=2,0,0,0,0,6 | -4.3 (0.47) |  |  |  |  | 3.6 (9.08)

18. Primary Outcome: Change From Baseline in PR Interval, QRS Interval, QT Interval and QT Interval Corrected by Fridericia's Formula (QTcF) Interval
Description: 12-lead ECG were performed in a supine position using an automated ECG machine that calculated PR interval, QRS interval, QT interval and QTcF interval. ECG measurements were performed in triplicate. When multiple ECGs were performed at the same planned timepoint, the average value of each parameter was used. Baseline was defined as latest pre-dose assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at 2 and 8 hours on Day 1; Days 2, 3, 4 and 5; Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32, 36 and 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Milliseconds
  PR Interval,2 hours Day1,n=12,6,5,9,8,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 8 | 6
  PR Interval,2 hours Day1,n=12,6,5,9,8,6 | -4.5 (9.46) | 3.9 (2.85) | 3.5 (8.47) | -4.3 (9.10) | 3.7 (1.075) | -7.5 (12.23)
  PR Interval,8 hours Day1,n=12,6,6,9,9,6 | -4.1 (8.49) | 3.1 (6.02) | -1.8 (3.72) | -4.5 (11.76) | 1.9 (11.39) | -3.3 (10.88)
  PR Interval,Day 2,n=12,6,6,9,9,6 | -2.7 (11.51) | 2.0 (4.11) | 1.4 (3.95) | -4.4 (9.86) | 6.2 (11.05) | -4.1 (11.25)
  PR Interval, Day 3,n=12,6,6,9,9,6 | 2.3 (6.68) | 5.2 (4.29) | 0.5 (5.62) | -3.6 (11.96) | 6.0 (7.60) | -1.4 (8.82)
  PR Interval,Day 4,n=12,6,6,9,9,6 | -0.6 (6.80) | 8.1 (5.21) | -2.5 (6.12) | -2.3 (8.88) | 8.6 (10.17) | -4.3 (7.54)
  PR Interval,Day 5,n=12,6,6,9,9,6 | 1.3 (6.22) | 8.3 (8.22) | 3.5 (10.05) | -0.2 (4.54) | 10.0 (8.44) | -1.2 (4.91)
  PR Interval,Week 1,n=12,6,6,9,9,6 | -0.3 (8.12) | 0.8 (5.58) | 2.2 (5.69) | -3.2 (12.26) | 7.0 (6.62) | 4.5 (6.73)
  PR Interval,Week 2,n=12,6,6,9,9,6 | -1.0 (8.62) | 5.3 (6.60) | 5.5 (10.34) | 1.8 (12.19) | 2.0 (12.64) | 1.0 (2.97)
  PR Interval,Week 4,n=12,6,6,8,9,6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 9 | 6
  PR Interval,Week 4,n=12,6,6,8,9,6 | 1.7 (10.27) | 5.2 (3.37) | 1.8 (12.71) | -1.8 (15.25) | 3.9 (11.28) | -4.0 (17.49)
  PR Interval,Week 8,n=12,6,6,9,9,6 | -3.1 (8.27) | 3.2 (9.65) | -2.6 (10.27) | -3.6 (10.33) | 3.4 (8.10) | -1.9 (9.55)
  PR Interval,Week 12,n=12,6,6,9,9,6 | -2.4 (7.87) | 3.9 (10.53) | -4.4 (12.18) | -3.8 (13.26) | 9.4 (8.33) | -2.1 (10.04)
  PR Interval,Week 18,n=12,6,6,9,9,6 | 1.5 (10.74) | 1.5 (3.99) | 0.1 (7.74) | -5.6 (11.87) | 7.3 (13.34) | -2.0 (9.72)
  PR Interval,Week 24,n=12,6,6,9,9,6 | 2.3 (7.98) | 1.4 (3.91) | 3.7 (7.25) | -7.4 (11.56) | 5.5 (12.45) | -5.6 (7.87)
  PR Interval,Week 26,n=12,6,6,9,9,6 | 1.1 (6.20) | 3.0 (4.67) | 3.7 (11.62) | -3.2 (13.01) | 6.9 (11.36) | -4.8 (11.69)
  PR Interval,Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  PR Interval,Week 32,n=6,6,6,0,0,6 | -4.3 (8.16) | 5.4 (7.23) | 0.0 (7.99) |  |  | -3.3 (11.91)
  PR Interval,Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  PR Interval,Week 36,n=6,0,0,9,9,0 | -0.5 (8.26) |  |  | -3.7 (8.49) | 2.9 (12.08) |
  PR Interval,Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  PR Interval,Week 40,n=2,0,0,0,0,6 | -13.7 (6.60) |  |  |  |  | -3.6 (8.56)
  QRS Interval,2 hours Day1,n=12,6,5,9,8,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 8 | 6
  QRS Interval,2 hours Day1,n=12,6,5,9,8,6 | 1.1 (4.87) | 0.2 (4.63) | -7.2 (4.97) | 0.0 (4.43) | -1.5 (6.14) | -1.2 (3.62)
  QRS Interval,8 hours Day1,n=12,6,6,9,9,6 | -0.3 (6.83) | -0.2 (6.81) | -4.0 (6.18) | -1.1 (3.18) | -2.8 (5.03) | -3.1 (4.42)
  QRS Interval,Day 2,n=12,6,6,9,9,6 | 1.8 (4.64) | 0.5 (4.63) | -4.9 (4.60) | -2.7 (5.28) | -3.0 (6.27) | -3.7 (4.62)
  QRS Interval, Day 3,n=12,6,6,9,9,6 | 1.4 (3.44) | 1.4 (4.18) | -1.3 (3.14) | -0.6 (4.03) | -2.6 (5.15) | -2.6 (1.54)
  QRS Interval,Day 4,n=12,6,6,9,9,6 | 0.4 (3.78) | 1.9 (3.72) | -7.8 (5.52) | 1.1 (5.28) | -0.7 (5.24) | -2.2 (3.38)
  QRS Interval,Day 5,n=12,6,6,9,9,6 | -0.5 (4.05) | 0.2 (5.85) | -7.3 (4.79) | -0.2 (5.40) | 0.7 (5.09) | -2.9 (2.35)
  QRS Interval,Week 1,n=12,6,6,9,9,6 | 2.3 (5.05) | 0.6 (5.85) | -3.7 (6.18) | 0.6 (4.90) | -2.4 (5.61) | -2.8 (4.20)
  QRS Interval,Week 2,n=12,6,6,9,9,6 | 2.1 (3.76) | 2.1 (4.82) | -3.9 (4.76) | 0.9 (2.86) | -3.0 (5.47) | -1.4 (3.11)
  QRS Interval,Week 4,n=12,6,6,8,9,6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 9 | 6
  QRS Interval,Week 4,n=12,6,6,8,9,6 | 2.0 (6.49) | 1.8 (7.34) | -6.5 (7.76) | 1.9 (4.79) | -2.6 (4.98) | -3.3 (3.39)
  QRS Interval,Week 8,n=12,6,6,9,9,6 | 1.9 (7.27) | -1.0 (4.35) | -3.6 (5.23) | 0.9 (4.12) | 0.5 (5.71) | -1.9 (1.83)
  QRS Interval,Week 12,n=12,6,6,9,9,6 | 1.6 (4.20) | 3.1 (3.28) | -4.4 (6.04) | -0.1 (5.23) | -2.5 (3.11) | -1.1 (3.21)
  QRS Interval,Week 18,n=12,6,6,9,9,6 | 0.6 (3.90) | 1.8 (2.79) | -5.0 (5.43) | 0.4 (3.16) | -2.9 (4.53) | -1.6 (4.17)
  QRS Interval,Week 24,n=12,6,6,9,9,6 | 0.6 (5.94) | 1.8 (6.53) | -6.5 (5.56) | -1.1 (3.76) | -3.1 (2.01) | -1.8 (5.12)
  QRS Interval,Week 26,n=12,6,6,9,9,6 | 0.0 (4.61) | 2.1 (4.64) | -5.5 (5.75) | 0.4 (5.55) | -2.7 (6.57) | 0.4 (3.40)
  QRS Interval,Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  QRS Interval,Week 32,n=6,6,6,0,0,6 | 2.9 (5.78) | 2.0 (5.17) | -6.1 (4.50) |  |  | -1.3 (2.56)
  QRS Interval,Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  QRS Interval,Week 36,n=6,0,0,9,9,0 | -3.7 (6.19) |  |  | 0.7 (5.14) | -3.9 (4.84) |
  QRS Interval,Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  QRS Interval,Week 40,n=2,0,0,0,0,6 | 0.0 (0.47) |  |  |  |  | -3.0 (3.47)
  QT Interval,2 hours Day1,n=12,6,5,9,8,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 8 | 6
  QT Interval,2 hours Day1,n=12,6,5,9,8,6 | -2.6 (22.55) | 14.8 (16.65) | 6.0 (11.28) | -2.9 (20.19) | -3.7 (23.95) | -9.2 (18.68)
  QT Interval,8 hours Day1,n=12,6,6,9,9,6 | -7.5 (16.46) | 6.7 (16.22) | 12.6 (18.53) | 1.5 (14.29) | -0.7 (29.93) | -7.6 (22.43)
  QT Interval,Day 2,n=12,6,6,9,9,6 | -4.9 (19.32) | 4.3 (14.01) | -14.1 (16.26) | -3.0 (18.80) | -6.1 (15.86) | -0.6 (11.09)
  QT Interval, Day 3,n=12,6,6,9,9,6 | -10.1 (19.82) | -0.9 (10.33) | -6.9 (14.95) | -7.6 (18.49) | -13.2 (15.20) | -2.4 (9.29)
  QT Interval,Day 4,n=12,6,6,9,9,6 | -12.3 (17.15) | -2.2 (14.32) | -15.9 (21.55) | -11.6 (25.81) | -10.9 (11.99) | -3.2 (17.05)
  QT Interval,Day 5,n=12,6,6,9,9,6 | -5.9 (14.18) | -2.2 (21.88) | -14.3 (13.83) | -9.5 (14.97) | -4.1 (18.72) | -1.3 (11.57)
  QT Interval,Week 1,n=12,6,6,9,9,6 | 5.3 (17.30) | 8.7 (14.19) | 0.0 (21.14) | -9.4 (19.82) | -1.0 (22.22) | -5.6 (23.13)
  QT Interval,Week 2,n=12,6,6,9,9,6 | 9.4 (16.23) | 12.9 (8.14) | 7.8 (17.65) | 1.0 (22.66) | -6.1 (17.10) | 8.3 (20.06)
  QT Interval,Week 4,n=12,6,6,8,9,6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 9 | 6
  QT Interval,Week 4,n=12,6,6,8,9,6 | 9.4 (20.43) | 11.0 (4.78) | -3.6 (24.50) | 3.3 (17.80) | 1.7 (34.52) | 14.0 (18.29)
  QT Interval,Week 8,n=12,6,6,9,9,6 | -0.6 (20.74) | 6.9 (9.28) | 1.0 (23.62) | 4.6 (19.06) | -2.0 (20.79) | 6.0 (15.76)
  QT Interval,Week 12,n=12,6,6,9,9,6 | -6.8 (20.64) | 8.1 (16.21) | 4.2 (22.53) | -6.5 (28.72) | -2.1 (26.69) | 1.1 (14.24)
  QT Interval,Week 18,n=12,6,6,9,9,6 | 7.3 (22.44) | 6.3 (15.00) | -2.8 (15.12) | -4.5 (19.10) | -6.7 (23.77) | 0.5 (12.14)
  QT Interval,Week 24,n=12,6,6,9,9,6 | 7.1 (23.22) | 4.2 (18.11) | -9.9 (27.45) | 0.7 (19.24) | -8.6 (19.00) | 7.9 (23.80)
  QT Interval,Week 26,n=12,6,6,9,9,6 | 2.3 (27.36) | 10.2 (12.92) | 0.9 (29.72) | -6.1 (22.91) | -9.8 (18.29) | 13.2 (20.96)
  QT Interval,Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  QT Interval,Week 32,n=6,6,6,0,0,6 | 5.7 (20.32) | 12.9 (12.12) | -14.4 (17.64) |  |  | 5.3 (14.64)
  QT Interval,Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  QT Interval,Week 36,n=6,0,0,9,9,0 | -6.4 (41.25) |  |  | -3.4 (29.83) | -9.3 (16.00) |
  QT Interval,Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  QT Interval,Week 40,n=2,0,0,0,0,6 | 23.5 (17.68) |  |  |  |  | -0.9 (24.13)
  QTcF Interval,2 hours Day1,n=12,6,5,9,8,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 8 | 6
  QTcF Interval,2 hours Day1,n=12,6,5,9,8,6 | -0.6 (9.11) | 4.1 (8.67) | -5.5 (8.11) | -3.4 (6.40) | -2.3 (5.38) | 6.4 (5.17)
  QTcF Interval,8 hours Day1,n=12,6,6,9,9,6 | -6.8 (12.97) | 4.3 (7.93) | -3.6 (12.32) | -1.4 (9.87) | -0.4 (8.32) | 2.1 (13.97)
  QTcF Interval,Day 2,n=12,6,6,9,9,6 | -4.0 (11.78) | 2.6 (8.43) | -12.8 (10.87) | -6.9 (9.34) | -5.9 (5.70) | -0.2 (10.66)
  QTcF Interval, Day 3,n=12,6,6,9,9,6 | -6.8 (14.99) | 0.4 (5.82) | -6.5 (9.14) | -5.3 (9.95) | -6.3 (10.71) | 1.9 (14.28)
  QTcF Interval,Day 4,n=12,6,6,9,9,6 | -4.9 (14.08) | 0.7 (7.62) | -6.1 (7.10) | -7.7 (12.56) | -4.8 (10.75) | 3.5 (17.05)
  QTcF Interval,Day 5,n=12,6,6,9,9,6 | -1.7 (11.97) | 1.5 (14.24) | -13.6 (11.17) | -4.7 (9.86) | -4.4 (14.31) | 3.9 (16.06)
  QTcF Interval,Week 1,n=12,6,6,9,9,6 | -0.2 (10.95) | 10.3 (7.33) | -6.7 (12.72) | -5.4 (8.38) | 2.8 (12.12) | 5.5 (13.80)
  QTcF Interval,Week 2,n=12,6,6,9,9,6 | 0.9 (16.40) | 6.3 (6.98) | -8.3 (8.21) | 3.7 (19.35) | -2.3 (12.64) | 11.5 (12.63)
  QTcF Interval,Week 4,n=12,6,6,8,9,6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 9 | 6
  QTcF Interval,Week 4,n=12,6,6,8,9,6 | -0.6 (11.22) | 7.3 (7.10) | -6.6 (20.63) | 0.5 (10.86) | -0.7 (10.97) | 11.4 (6.33)
  QTcF Interval,Week 8,n=12,6,6,9,9,6 | -2.8 (13.76) | 5.2 (9.28) | -4.8 (14.70) | -1.7 (11.96) | -2.9 (14.10) | 8.1 (20.96)
  QTcF Interval,Week 12,n=12,6,6,9,9,6 | -6.4 (14.39) | 5.9 (13.50) | -5.3 (10.66) | -5.9 (10.93) | -1.1 (11.91) | 4.7 (10.23)
  QTcF Interval,Week 18,n=12,6,6,9,9,6 | -0.5 (11.73) | 4.8 (6.79) | -10.4 (9.42) | -0.6 (12.29) | -5.2 (12.81) | 5.9 (11.16)
  QTcF Interval,Week 24,n=12,6,6,9,9,6 | 1.4 (15.42) | 3.0 (10.83) | -7.2 (12.14) | 0.4 (7.96) | -3.9 (12.69) | 10.1 (15.15)
  QTcF Interval,Week 26,n=12,6,6,9,9,6 | -1.9 (16.58) | 9.6 (9.37) | -3.9 (14.54) | -1.7 (10.65) | -4.4 (12.21) | 12.8 (8.59)
  QTcF Interval,Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  QTcF Interval,Week 32,n=6,6,6,0,0,6 | 0.4 (10.98) | 1.3 (7.93) | -13.8 (8.76) |  |  | 11.7 (13.74)
  QTcF Interval,Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  QTcF Interval,Week 36,n=6,0,0,9,9,0 | -3.7 (24.89) |  |  | -4.3 (13.45) | -5.5 (14.23) |
  QTcF Interval,Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  QTcF Interval,Week 40,n=2,0,0,0,0,6 | 12.0 (17.44) |  |  |  |  | 7.5 (14.62)

19. Secondary Outcome: Area Under the Curve From Time Zero to Infinity (AUC[0-inf]) of GSK3511294 2 mg and 10 mg
Description: Blood samples were collected from participants at indicated time points and analyzed for AUC (0-inf). Pharmacokinetic parameters were calculated by standard non compartmental analysis. Pharmacokinetic Population included participants in the Safety population for whom a pharmcokinetic sample was obtained and analyzed.
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, and 26 post-dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*microgram per milliliter
Arm/Group | GSK3511294 2mg | GSK3511294 10mg
Number analyzed (Participants) | 6 | 6
Day*microgram per milliliter | 24.795 (51.6) | 68.904 (23.6)

20. Secondary Outcome: AUC(0-inf) of GSK3511294 30 mg and 100 mg
Description: Blood samples were collected from participants at indicated time points and analyzed for AUC (0-inf). Pharmacokinetic parameters were calculated by standard non compartmental analysis.
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, 26 and 36 post-dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*microgram per milliliter
Arm/Group | GSK3511294 30mg | GSK3511294 100mg
Number analyzed (Participants) | 9 | 9
Day*microgram per milliliter | 208.308 (39.6) | 846.686 (7.3)

21. Secondary Outcome: AUC(0-inf) of GSK3511294 300 mg
Description: as for outcome 20
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32 and 40 post-dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*microgram per milliliter
Arm/Group | GSK3511294 300mg
Number analyzed (Participants) | 6
Day*microgram per milliliter | 1873.657 (25.5)

22. Secondary Outcome: Area Under the Curve From Time Zero to the Last Measurable Concentration (AUC[0-t]) of GSK3511294 2 mg and 10 mg
Description: Blood samples were collected from participants at indicated time points and analyzed for AUC (0-t). Pharmacokinetic parameters were calculated by standard non compartmental analysis.
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, and 26 post-dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*microgram per milliliter
Arm/Group | GSK3511294 2mg | GSK3511294 10mg
Number analyzed (Participants) | 6 | 6
Day*microgram per milliliter | 18.369 (59.2) | 62.101 (28.4)

23. Secondary Outcome: AUC(0-t) of GSK3511294 30 mg and 100 mg
Description: as for outcome 22
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, 26 and 36 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*microgram per milliliter
Arm/Group | GSK3511294 30mg | GSK3511294 100mg
Number analyzed (Participants) | 9 | 9
Day*microgram per milliliter | 201.434 (41.1) | 830.245 (7.4)

24. Secondary Outcome: AUC(0-t) of GSK3511294 300 mg
Description: Blood samples were collected from participants at indicated time points and analyzed for AUC (0-t). Pharmacokinetic parameters was calculated by standard non compartmental analysis.
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32 and 40 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*microgram per milliliter
Arm/Group | GSK3511294 300mg
Number analyzed (Participants) | 6
Day*microgram per milliliter | 1855.619 (25.8)

25. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Week 4 (AUC[0-Week 4]) of GSK3511294
Description: Blood samples were collected from participants at indicated time points and analyzed for AUC (0-Week 4). Pharmacokinetic parameters was calculated by standard non compartmental analysis.
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, and 4 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*microgram per milliliter
Arm/Group | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 6 | 6 | 9 | 9 | 6
Day*microgram per milliliter | 6.856 (22.0) | 19.685 (14.0) | 62.994 (40.6) | 292.698 (11.0) | 676.055 (22.7)

26. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Week 12 (AUC[0-Week 12]) of GSK3511294
Description: Blood samples were collected from participants at indicated time points and analyzed for AUC (0-Week 12). Pharmacokinetic parameters were calculated by standard non compartmental analysis.
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8 and 12 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*microgram per milliliter
Arm/Group | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 6 | 6 | 9 | 9 | 6
Day*microgram per milliliter | 16.102 (37.1) | 48.389 (22.7) | 148.798 (37.8) | 663.984 (8.1) | 1445.726 (23.8)

27. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Week 26 (AUC [0-Week 26]) of GSK3511294
Description: Blood samples were collected from participants at indicated time points and analyzed for AUC (0-Week 26). Pharmacokinetic parameters was calculated by standard non compartmental analysis.
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24 and 26 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*microgram per milliliter
Arm/Group | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 6 | 6 | 9 | 9 | 6
Day*microgram per milliliter | 21.829 (42.7) | 64.453 (24.3) | 199.893 (39.9) | 805.359 (7.7) | 1789.451 (26.3)

28. Secondary Outcome: Percentage of AUC (0-inf) Obtained by Extrapolation (%AUCex) of GSK3511294 2 mg and 10 mg
Description: Blood samples were collected from participants at indicated time points and analyzed for %AUCex. Pharmacokinetic parameters was calculated by standard non compartmental analysis.
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, and 26 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUCex
Arm/Group | GSK3511294 2mg | GSK3511294 10mg
Number analyzed (Participants) | 6 | 6
Percentage of AUCex | 24.3560 (35.8) | 7.7705 (81.6)

29. Secondary Outcome: %AUCex of GSK3511294 30 mg and 100 mg
Description: as for outcome 28
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, 26 and 36 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUCex
Arm/Group | GSK3511294 30mg | GSK3511294 100mg
Number analyzed (Participants) | 9 | 9
Percentage of AUCex | 2.9636 (55.6) | 1.4162 (88.3)

30. Secondary Outcome: %AUCex of GSK3511294 300 mg
Description: as for outcome 28
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32 and 40 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUCex
Arm/Group | GSK3511294 300mg
Number analyzed (Participants) | 6
Percentage of AUCex | 0.9096 (35.1)

31. Secondary Outcome: Maximum Observed Concentration (Cmax) of GSK3511294 2 mg and 10 mg
Description: Blood samples were collected from participants at indicated time points and analyzed for Cmax. Pharmacokinetic parameters was calculated by standard non compartmental analysis.
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, and 26 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | GSK3511294 2mg | GSK3511294 10mg
Number analyzed (Participants) | 6 | 6
Microgram per milliliter | 0.3400 (25.3) | 0.8759 (18.3)

32. Secondary Outcome: Cmax of GSK3511294 30 mg and 100 mg
Description: as for outcome 31
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, 26 and 36 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | GSK3511294 30mg | GSK3511294 100mg
Number analyzed (Participants) | 9 | 9
Microgram per milliliter | 2.8101 (41.1) | 12.2471 (15.9)

33. Secondary Outcome: Cmax of GSK3511294 300 mg
Description: as for outcome 31
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32 and 40 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | GSK3511294 300mg
Number analyzed (Participants) | 6
Microgram per milliliter | 28.5987 (23.3)

34. Secondary Outcome: Time of Occurrence of Cmax (Tmax) of GSK3511294 2 mg and 10 mg
Description: Blood samples were collected from participants at indicated time points and analyzed for Tmax. Pharmacokinetic parameters was calculated by standard non compartmental analysis.
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, and 26 post-dose
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Days
Arm/Group | GSK3511294 2mg | GSK3511294 10mg
Number analyzed (Participants) | 6 | 6
Days | 10.966 [6.99 to 27.98] | 7.956 [7.00 to 28.91]

35. Secondary Outcome: Tmax of GSK3511294 30 mg and 100 mg
Description: as for outcome 34
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, 26 and 36 post-dose
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Days
Arm/Group | GSK3511294 30mg | GSK3511294 100mg
Number analyzed (Participants) | 9 | 9
Days | 13.943 [4.00 to 28.02] | 13.970 [3.97 to 16.00]

36. Secondary Outcome: Tmax of GSK3511294 300 mg
Description: as for outcome 34
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32 and 40 post-dose
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Days
Arm/Group | GSK3511294 300mg
Number analyzed (Participants) | 6
Days | 13.909 [2.00 to 15.00]

37. Secondary Outcome: Time of Last Quantifiable Concentration (Tlast) of GSK3511294 2 mg and 10 mg
Description: Blood samples were collected from participants at indicated time points and analyzed for Tlast. Pharmacokinetic parameters was calculated by standard non compartmental analysis.
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, and 26 post-dose
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Days
Arm/Group | GSK3511294 2mg | GSK3511294 10mg
Number analyzed (Participants) | 6 | 6
Days | 84.47 [84.0 to 182.0] | 176.46 [126.0 to 185.0]

38. Secondary Outcome: Tlast of GSK3511294 30 mg and 100 mg
Description: as for outcome 37
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, 26 and 36 post-dose
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Days
Arm/Group | GSK3511294 30mg | GSK3511294 100mg
Number analyzed (Participants) | 9 | 9
Days | 182.01 [182.0 to 254.8] | 252.00 [250.0 to 255.0]

39. Secondary Outcome: Tlast of GSK3511294 300 mg
Description: as for outcome 37
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32 and 40 post-dose
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Days
Arm/Group | GSK3511294 300mg
Number analyzed (Participants) | 6
Days | 279.99 [278.0 to 283.0]

40. Secondary Outcome: Apparent Clearance Following Subcutaneous Dosing (CL/F) of GSK3511294 2 mg and 10 mg
Description: Blood samples were collected from participants at indicated time points and analyzed for CL/F. CL/F was calculated as dose divided by AUC(0-inf). Pharmacokinetic parameters was calculated by standard non compartmental analysis.
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, and 26 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per day
Arm/Group | GSK3511294 2mg | GSK3511294 10mg
Number analyzed (Participants) | 6 | 6
Liters per day | 0.08066 (51.6) | 0.14513 (23.6)

41. Secondary Outcome: CL/F of GSK3511294 30 mg and 100 mg
Description: as for outcome 40
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, 26 and 36 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per day
Arm/Group | GSK3511294 30mg | GSK3511294 100mg
Number analyzed (Participants) | 9 | 9
Liters per day | 0.14402 (39.6) | 0.11811 (7.3)

42. Secondary Outcome: CL/F of GSK3511294 300 mg
Description: as for outcome 40
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32 and 40 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per day
Arm/Group | GSK3511294 300mg
Number analyzed (Participants) | 6
Liters per day | 0.16011 (25.5)

43. Secondary Outcome: Apparent Volume of Distribution After Subcutaneous Administration (Vd/F) of GSK3511294 2 mg and 10 mg
Description: Blood samples were collected from participants at indicated time points and analyzed for Vd/F. Vd/F was calculated as dose divided by terminal elimination rate constant (lambda_z) *AUC(0-inf). Pharmacokinetic parameters were calculated by standard non compartmental analysis.
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, and 26 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | GSK3511294 2mg | GSK3511294 10mg
Number analyzed (Participants) | 6 | 6
Liters | 6.113 (37.6) | 9.193 (34.7)

44. Secondary Outcome: Vd/F of GSK3511294 30 mg and 100 mg
Description: Blood samples were collected from participants at indicated time points and analyzed for Vd/F. Vd/F was calculated as dose divided by [lambda_z *AUC(0-inf)]. Pharmacokinetic parameters was calculated by standard non compartmental analysis.
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, 26 and 36 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | GSK3511294 30mg | GSK3511294 100mg
Number analyzed (Participants) | 9 | 9
Liters | 7.812 (40.4) | 6.630 (12.1)

45. Secondary Outcome: Vd/F of GSK3511294 300 mg
Description: as for outcome 44
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32 and 40 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | GSK3511294 300mg
Number analyzed (Participants) | 6
Liters | 9.337 (30.6)

46. Secondary Outcome: Terminal Phase Elimination Rate Constant (Lambda_z) of GSK3511294 2 mg and 10 mg
Description: Blood samples were collected from participants at indicated time points and analyzed for lambda_z. Pharmacokinetic parameters was calculated by standard non compartmental analysis.
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, and 26 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day^-1
Arm/Group | GSK3511294 2mg | GSK3511294 10mg
Number analyzed (Participants) | 6 | 6
Day^-1 | 0.013195 (37.3) | 0.015787 (16.2)

47. Secondary Outcome: Lambda_z of GSK3511294 30 mg and 100 mg
Description: as for outcome 46
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, 26 and 36 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day^-1
Arm/Group | GSK3511294 30mg | GSK3511294 100mg
Number analyzed (Participants) | 9 | 9
Day^-1 | 0.018435 (10.7) | 0.017813 (11.7)

48. Secondary Outcome: Lambda_z of GSK3511294 300 mg
Description: as for outcome 46
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32 and 40 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day^-1
Arm/Group | GSK3511294 300mg
Number analyzed (Participants) | 6
Day^-1 | 0.017148 (6.3)

49. Secondary Outcome: Terminal Phase Half-life (t1/2) of GSK3511294 2 mg and 10 mg
Description: Blood samples were collected from participants at indicated time points and analyzed for t1/2. Pharmacokinetic parameters was calculated by standard non compartmental analysis.
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, and 26 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | GSK3511294 2mg | GSK3511294 10mg
Number analyzed (Participants) | 6 | 6
Days | 52.531 (37.3) | 43.907 (16.2)

50. Secondary Outcome: T1/2 of GSK3511294 30 mg and 100 mg
Description: as for outcome 49
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, 26 and 36 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | GSK3511294 30mg | GSK3511294 100mg
Number analyzed (Participants) | 9 | 9
Days | 37.599 (10.7) | 38.913 (11.7)

51. Secondary Outcome: T1/2 of GSK3511294 300 mg
Description: as for outcome 49
Time Frame: Pre-dose, 2 and 8 hours on Day 1; Days 2,3,5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32 and 40 post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | GSK3511294 300mg
Number analyzed (Participants) | 6
Days | 40.422 (6.3)

52. Secondary Outcome: Ratio to Baseline in Absolute Blood Eosinophil Count
Description: Blood samples were collected at indicated time-points. Analysis was performed using a mixed model repeated measures analysis (MMRM) model on log-transformed data with fixed categorical effects of treatment, planned timepoint and treatment-by-planned timepoint interaction and fixed continuous covariates of log Baseline blood eosinophil count and log Baseline blood eosinophil count-by-planned timepoint interaction. Baseline is defined as the latest predose non-missing blood eosinophil count. Ratio to Baseline is defined as post-dose visit value divided by Baseline value. Pharmacodynamic Population included participants in the 'Safety' population for whom a post-dose pharmacodynamic (ie blood eosinophil) sample was obtained and analyzed.
Time Frame: Baseline, Days 2, 3, 4, 5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32, 36, and 40
Population: Pharmacodynamic Population. Only those participants with planned assessments at that particular time point has been presented (represented by n=X in category titles)
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio of eosinophils in blood
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Ratio of eosinophils in blood
  Day 2, n=12, 6, 6, 8, 9, 6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 9 | 6
  Day 2, n=12, 6, 6, 8, 9, 6 | 1.083 [0.828 to 1.418] | 0.562 [0.382 to 0.827] | 0.522 [0.356 to 0.765] | 0.434 [0.313 to 0.601] | 0.496 [0.364 to 0.677] | 0.466 [0.317 to 0.683]
  Day 3, n=12, 6, 6, 9, 9, 6 | 0.977 [0.747 to 1.279] | 0.431 [0.293 to 0.633] | 0.350 [0.238 to 0.512] | 0.281 [0.205 to 0.386] | 0.262 [0.192 to 0.357] | 0.403 [0.275 to 0.591]
  Day 4, n=12, 6, 6, 8, 8, 6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 8 | 6
  Day 4, n=12, 6, 6, 8, 8, 6 | 1.008 [0.770 to 1.319] | 0.400 [0.272 to 0.589] | 0.340 [0.232 to 0.499] | 0.215 [0.155 to 0.298] | 0.250 [0.182 to 0.344] | 0.360 [0.246 to 0.528]
  Day 5, n=11, 6, 6, 9, 9, 6: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 6
  Day 5, n=11, 6, 6, 9, 9, 6 | 0.927 [0.705 to 1.220] | 0.300 [0.204 to 0.442] | 0.267 [0.182 to 0.391] | 0.219 [0.159 to 0.300] | 0.280 [0.205 to 0.382] | 0.299 [0.204 to 0.438]
  Week 1, n=12, 6, 6, 9, 9, 5: number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 5
  Week 1, n=12, 6, 6, 9, 9, 5 | 1.136 [0.868 to 1.487] | 0.304 [0.206 to 0.447] | 0.223 [0.152 to 0.326] | 0.226 [0.165 to 0.311] | 0.237 [0.173 to 0.323] | 0.250 [0.167 to 0.373]
  Week 2, n=12, 6, 5, 9, 9, 6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Week 2, n=12, 6, 5, 9, 9, 6 | 1.174 [0.897 to 1.536] | 0.274 [0.186 to 0.403] | 0.225 [0.151 to 0.336] | 0.170 [0.124 to 0.233] | 0.214 [0.157 to 0.292] | 0.265 [0.180 to 0.388]
  Week 4,n=12, 6, 5, 9, 9, 6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Week 4,n=12, 6, 5, 9, 9, 6 | 1.062 [0.812 to 1.390] | 0.198 [0.134 to 0.291] | 0.195 [0.131 to 0.290] | 0.131 [0.095 to 0.179] | 0.185 [0.135 to 0.252] | 0.180 [0.123 to 0.264]
  Week 8, n=12, 6, 6, 9, 9, 6 | 1.095 [0.837 to 1.434] | 0.201 [0.137 to 0.296] | 0.129 [0.088 to 0.189] | 0.102 [0.075 to 0.140] | 0.126 [0.092 to 0.172] | 0.178 [0.121 to 0.261]
  Week 12, n=12, 5, 6, 9, 9, 5: number analyzed (Participants) | 12 | 5 | 6 | 9 | 9 | 5
  Week 12, n=12, 5, 6, 9, 9, 5 | 1.031 [0.788 to 1.350] | 0.373 [0.250 to 0.557] | 0.171 [0.116 to 0.250] | 0.123 [0.089 to 0.168] | 0.161 [0.118 to 0.220] | 0.164 [0.110 to 0.244]
  Week 18, n=12, 6, 6, 9, 9, 6 | 1.079 [0.824 to 1.412] | 0.466 [0.317 to 0.685] | 0.314 [0.214 to 0.460] | 0.152 [0.111 to 0.208] | 0.139 [0.102 to 0.190] | 0.179 [0.122 to 0.262]
  Week 24, n=11, 6, 6, 9, 9, 6: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 6
  Week 24, n=11, 6, 6, 9, 9, 6 | 1.005 [0.763 to 1.322] | 0.661 [0.449 to 0.972] | 0.563 [0.384 to 0.825] | 0.285 [0.208 to 0.391] | 0.149 [0.109 to 0.203] | 0.202 [0.137 to 0.296]
  Week 26, n=12, 6, 6, 9, 9, 6 | 1.119 [0.855 to 1.464] | 0.776 [0.527 to 1.141] | 0.663 [0.452 to 0.972] | 0.317 [0.231 to 0.435] | 0.199 [0.146 to 0.271] | 0.186 [0.127 to 0.273]
  Week 32, n=6, 6, 6, 0, 0, 6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Week 32, n=6, 6, 6, 0, 0, 6 | 0.912 [0.656 to 1.268] | 0.968 [0.655 to 1.430] | 0.837 [0.569 to 1.229] |  |  | 0.210 [0.142 to 0.308]
  Week 36, n=6, 0, 0, 9, 9, 0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Week 36, n=6, 0, 0, 9, 9, 0 | 0.975 [0.691 to 1.376] |  |  | 0.858 [0.624 to 1.180] | 0.374 [0.274 to 0.511] |
  Week 40, n=2, 0, 0, 0, 0, 6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Week 40, n=2, 0, 0, 0, 0, 6 | 1.210 [0.604 to 2.422] |  |  |  |  | 0.258 [0.172 to 0.387]

53. Secondary Outcome: Number of Participants With Anti-drug Antibody (ADA) Binding to GSK3511294
Description: Serum samples were collected to determine the presence of anti-GSK3511294 binding antibodies using a validated bioanalytical method. Data for any time post-Baseline is reported. The results were categorized as negative, transient positive (defined as a single confirmatory positive immunogenic response that does not occur at the final study assessment) and persistent positive (defined as a confirmatory positive immunogenic response for at least 2 consecutive assessments or a single result at the final study assessment).
Time Frame: Up to Week 40
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Participants
  Negative | 12 | 6 | 5 | 4 | 7 | 5
  Transient positive | 0 | 0 | 0 | 0 | 1 | 0
  Persistent positive | 0 | 0 | 1 | 5 | 1 | 1

54. Secondary Outcome: Titers of Binding ADA to GSK3511294
Description: Serum samples were collected to determine the presence of anti-GSK3511294 binding antibodies using a validated bioanalytical method. Data for any time post-Baseline is reported. Titer was only measured when a positive result was found.
Time Frame: Up to Week 40
Population: Safety Population. Only participants with positive results for ADA were analyzed.
Measure: Median (Full Range); unit: Titer
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 0 | 0 | 1 | 5 | 2 | 1
Titer |  |  | 80.0 [80 to 80] | 160.0 [80 to 320] | 80.0 [80 to 80] | 80.0 [80 to 320]

55. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters Like Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), and Aspartate Aminotransferase (AST)
Description: Blood samples were collected at indicated time-points for analysis of clinical parameters like ALP, AST and ALT. Baseline was defined as latest pre-dose assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 2, 3, 4 and 5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32, 36 and 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
International units per Liter
  ALT, Day 2,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  ALT, Day 2,n=12,6,5,9,9,6 | -0.3 (5.12) | 0.3 (3.56) | 4.0 (14.20) | -1.6 (2.07) | -0.1 (3.26) | -0.7 (2.73)
  ALT, Day 3,n=12,6,6,9,9,6 | 0.3 (5.96) | 2.5 (8.17) | 5.3 (17.94) | -0.6 (2.51) | -1.0 (3.20) | 1.2 (4.96)
  ALT, Day 4,n=12,6,6,9,9,6 | 1.0 (5.85) | 3.3 (11.08) | 4.2 (13.83) | -1.2 (1.86) | -0.1 (2.71) | 1.2 (3.43)
  ALT, Day 5,n=12,6,6,9,9,6 | 1.7 (7.96) | 2.0 (9.74) | 2.3 (8.91) | -0.6 (3.64) | 0.2 (3.42) | 4.5 (5.32)
  ALT, Week 1,n=12,6,6,9,9,5: number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 5
  ALT, Week 1,n=12,6,6,9,9,5 | 1.2 (7.76) | 1.3 (5.92) | 2.8 (7.36) | 0.7 (3.61) | 0.6 (4.98) | 1.2 (5.54)
  ALT, Week 2,n=12,6,6,9,9,6 | -0.2 (5.57) | -5.3 (7.97) | -1.3 (4.32) | 0.3 (4.85) | -2.3 (4.97) | 3.0 (2.53)
  ALT, Week 4,n=12,6,6,9,9,6 | -0.3 (6.43) | -4.3 (7.63) | 0.7 (4.23) | 1.4 (9.41) | -2.6 (2.55) | -2.8 (4.36)
  ALT, Week 8,n=12,6,6,9,9,6 | 0.3 (7.25) | -3.3 (10.39) | 2.5 (6.53) | -1.6 (3.40) | 1.8 (9.56) | -3.0 (4.77)
  ALT, Week 12,n=12,6,6,9,9,6 | -0.9 (6.07) | -1.7 (4.18) | 0.5 (3.94) | -0.4 (1.94) | 3.0 (5.12) | -0.7 (2.66)
  ALT, Week 18,n=12,6,6,9,9,6 | -0.1 (6.13) | -3.5 (7.56) | 1.0 (10.30) | 1.9 (8.81) | 4.4 (6.93) | -0.7 (5.20)
  ALT, Week 24,n=12,6,6,9,9,6 | 0.3 (12.11) | -3.5 (7.64) | 5.2 (14.18) | 2.2 (10.76) | 7.3 (12.97) | 0.8 (5.34)
  ALT, Week 26,n=12,6,6,9,9,6 | -2.1 (6.13) | -0.8 (6.79) | -0.5 (6.47) | 5.1 (19.63) | 6.2 (13.08) | 2.5 (7.87)
  ALT, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  ALT, Week 32,n=6,6,6,0,0,6 | 1.5 (8.04) | -1.7 (9.89) | -1.0 (3.29) |  |  | -3.0 (4.60)
  ALT, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  ALT, Week 36,n=6,0,0,9,9,0 | 0.3 (8.29) |  |  | 1.3 (6.86) | 5.0 (7.84) |
  ALT, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  ALT, Week 40,n=2,0,0,0,0,6 | -3.5 (7.78) |  |  |  |  | 1.2 (8.08)
  AST, Day 2,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  AST, Day 2,n=12,6,5,9,9,6 | -3.5 (3.55) | -1.2 (2.48) | -0.8 (7.19) | -2.6 (4.28) | -3.9 (5.42) | -3.7 (3.88)
  AST, Day 3,n=12,6,6,9,9,6 | -3.8 (4.86) | -0.8 (4.62) | -1.2 (7.22) | -1.8 (3.80) | -5.6 (6.58) | -3.2 (4.79)
  AST, Day 4,n=12,6,6,9,9,6 | -4.3 (4.27) | -0.8 (5.08) | -2.0 (4.34) | -2.9 (2.93) | -4.9 (6.33) | -3.3 (4.93)
  AST, Day 5,n=12,6,6,9,9,6 | -2.6 (4.10) | -0.5 (5.28) | -1.7 (3.67) | -3.2 (3.31) | -3.7 (7.57) | -2.0 (5.83)
  AST, Week 1,n=12,6,6,9,9,5: number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 5
  AST, Week 1,n=12,6,6,9,9,5 | -2.8 (4.12) | 0.0 (3.74) | -0.2 (2.32) | -1.9 (2.85) | -3.3 (4.53) | -4.6 (4.39)
  AST, Week 2,n=12,6,6,9,9,6 | -1.5 (4.66) | -0.3 (4.55) | -2.5 (2.88) | 1.0 (9.19) | -3.8 (6.44) | -0.7 (4.80)
  AST, Week 4,n=12,6,6,9,9,6 | -1.5 (3.97) | -2.3 (3.83) | 0.0 (6.03) | 0.0 (4.90) | -4.3 (6.87) | -4.2 (5.91)
  AST, Week 8,n=12,6,6,9,9,6 | -0.9 (7.45) | -1.8 (3.66) | 0.5 (3.02) | -0.2 (3.77) | -1.0 (10.58) | -4.7 (4.50)
  AST, Week 12,n=12,6,6,9,9,6 | -2.8 (2.79) | -1.2 (1.94) | 1.2 (3.71) | -1.2 (2.17) | -1.4 (6.98) | -2.0 (5.83)
  AST, Week 18,n=12,6,6,9,9,6 | -1.8 (4.14) | -1.2 (2.86) | 1.3 (10.09) | -0.7 (3.64) | -1.8 (5.56) | -3.3 (5.61)
  AST, Week 24,n=12,6,6,9,9,6 | 1.2 (18.52) | 1.3 (2.73) | 0.8 (5.42) | -1.1 (5.64) | -2.8 (8.76) | -1.8 (3.06)
  AST, Week 26,n=12,6,6,9,9,6 | -2.7 (4.08) | 1.8 (1.60) | 0.2 (3.37) | 0.0 (7.00) | 0.1 (9.21) | 0.2 (3.97)
  AST, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  AST, Week 32,n=6,6,6,0,0,6 | -2.7 (3.39) | 0.5 (3.33) | -2.5 (1.52) |  |  | -3.5 (5.47)
  AST, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  AST, Week 36,n=6,0,0,9,9,0 | -1.0 (4.69) |  |  | -2.0 (4.36) | -3.2 (6.70) |
  AST, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  AST, Week 40,n=2,0,0,0,0,6 | -7.5 (6.36) |  |  |  |  | 3.0 (13.24)
  ALP, Day 2,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  ALP, Day 2,n=12,6,5,9,9,6 | -1.8 (4.84) | -3.3 (1.37) | 1.0 (4.18) | -4.9 (2.80) | 1.3 (7.28) | -1.5 (7.77)
  ALP, Day 3,n=12,6,6,9,9,6 | -1.8 (5.66) | -2.7 (2.94) | 0.3 (8.52) | -1.8 (3.99) | -0.6 (5.32) | 0.2 (5.88)
  ALP, Day 4,n=12,6,6,9,9,6 | -1.7 (5.30) | -1.3 (3.20) | 0.0 (9.17) | -1.9 (3.62) | -0.2 (6.34) | -1.3 (6.09)
  ALP, Day 5,n=12,6,6,9,9,6 | 0.1 (5.74) | -2.0 (3.52) | 0.3 (4.76) | -1.4 (5.25) | 1.9 (9.44) | -1.2 (5.12)
  ALP, Week 1,n=12,6,6,9,9,5: number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 5
  ALP, Week 1,n=12,6,6,9,9,5 | 0.2 (5.86) | -2.2 (5.56) | -2.5 (6.06) | -0.7 (6.18) | -1.1 (4.62) | -1.2 (7.53)
  ALP, Week 2,n=12,6,6,9,9,6 | 1.0 (3.44) | -8.2 (6.52) | -4.2 (3.54) | -0.6 (3.91) | 3.1 (5.25) | -1.0 (8.32)
  ALP, Week 4,n=12,6,6,9,9,6 | 1.4 (4.81) | -8.2 (8.30) | -1.2 (3.97) | -3.2 (4.32) | 2.6 (5.50) | -2.2 (7.81)
  ALP, Week 8,n=12,6,6,9,9,6 | 1.9 (6.88) | -2.0 (4.82) | 1.0 (10.06) | -4.4 (4.03) | 3.7 (3.61) | -0.8 (8.30)
  ALP, Week 12,n=12,6,6,9,9,6 | -0.6 (6.43) | -4.3 (7.09) | 7.2 (10.46) | -2.8 (2.82) | 3.1 (11.58) | -0.3 (5.09)
  ALP, Week 18,n=12,6,6,9,9,6 | 3.1 (6.82) | -2.0 (6.48) | -1.7 (4.84) | 1.9 (6.79) | 3.8 (8.27) | -3.5 (6.80)
  ALP, Week 24,n=12,6,6,9,9,6 | 3.8 (12.21) | -1.2 (7.94) | -1.0 (4.73) | 1.2 (10.51) | 5.8 (8.39) | -0.7 (6.74)
  ALP, Week 26,n=12,6,6,9,9,6 | 3.2 (8.64) | -6.2 (8.30) | -2.2 (4.02) | 0.4 (10.75) | 4.8 (8.24) | -1.7 (6.02)
  ALP, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  ALP, Week 32,n=6,6,6,0,0,6 | -2.0 (8.51) | -3.3 (8.50) | 0.2 (5.31) |  |  | -1.0 (7.72)
  ALP, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  ALP, Week 36,n=6,0,0,9,9,0 | 9.0 (15.57) |  |  | -0.6 (11.19) | 7.2 (8.39) |
  ALP, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  ALP, Week 40,n=2,0,0,0,0,6 | -5.5 (0.71) |  |  |  |  | -3.7 (9.48)

56. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter Like Glucose, Calcium, Potassium, Sodium, Blood Urea Nitrogen (BUN), and Magnesium
Description: Blood samples were collected at indicated time-points for analysis of clinical parameters like glucose, calcium, potassium, sodium, BUN, and magnesium. Baseline was defined as latest pre-dose assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 2, 3, 4 and 5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32, 36 and 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Millimoles per liter
  Glucose, Day 2,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Glucose, Day 2,n=12,6,5,9,9,6 | 0.06 (0.912) | -0.13 (0.418) | 0.14 (0.439) | -0.11 (0.533) | -0.72 (0.948) | 0.20 (0.352)
  Glucose, Day 3,n=12,6,6,9,9,6 | -0.28 (0.673) | -0.10 (1.215) | -0.93 (1.117) | -0.18 (0.455) | -0.21 (0.647) | 0.15 (0.521)
  Glucose, Day 4,n=12,6,6,9,9,6 | -0.11 (0.712) | 0.12 (0.987) | -0.33 (0.857) | 0.26 (0.940) | -0.34 (1.364) | 0.50 (1.103)
  Glucose, Day 5,n=12,6,6,9,9,6 | -0.06 (0.647) | -0.07 (0.612) | 0.28 (0.958) | 0.01 (0.775) | -0.17 (0.728) | 0.05 (0.539)
  Glucose, Week 1,n=11,6,6,9,9,5: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 5
  Glucose, Week 1,n=11,6,6,9,9,5 | 0.00 (0.656) | -0.35 (0.394) | -0.18 (1.280) | -0.20 (0.624) | -0.23 (1.015) | 0.50 (1.345)
  Glucose, Week 2,n=12,6,6,9,9,6 | 0.03 (0.396) | -0.05 (0.295) | 0.00 (0.525) | -0.02 (1.027) | -0.18 (0.902) | -0.10 (0.155)
  Glucose, Week 4,n=12,6,6,9,9,6 | 0.19 (0.783) | -0.33 (0.543) | 0.03 (0.582) | -0.28 (0.678) | -0.08 (0.919) | 0.33 (0.476)
  Glucose, Week 8,n=12,6,6,9,9,6 | 0.06 (0.444) | -0.42 (0.585) | 0.27 (0.824) | 0.04 (0.430) | -0.36 (1.193) | 0.42 (0.722)
  Glucose, Week 12,n=12,6,6,9,9,6 | 0.32 (0.606) | -0.15 (0.428) | 0.13 (1.093) | 0.08 (0.905) | -0.66 (0.760) | 0.23 (0.432)
  Glucose, Week 18,n=12,6,6,9,9,6 | 0.03 (0.548) | -0.02 (0.331) | 0.42 (1.017) | -0.17 (0.541) | -0.23 (0.825) | 0.15 (0.288)
  Glucose, Week 24,n=12,6,6,9,9,6 | 0.38 (1.131) | -0.13 (0.333) | 0.02 (0.773) | -0.27 (0.654) | -0.26 (0.928) | 0.50 (0.590)
  Glucose, Week 26,n=12,6,6,9,9,6 | 0.18 (0.506) | -0.10 (0.346) | 0.62 (1.144) | -0.09 (0.362) | -0.22 (0.758) | 0.38 (0.445)
  Glucose, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Glucose, Week 32,n=6,6,6,0,0,6 | 0.40 (1.233) | 0.02 (0.194) | -0.28 (0.703) |  |  | 0.32 (0.354)
  Glucose, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Glucose, Week 36,n=6,0,0,9,9,0 | 0.17 (0.493) |  |  | -0.26 (0.436) | -0.07 (0.996) |
  Glucose, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Glucose, Week 40,n=2,0,0,0,0,6 | 0.40 (0.566) |  |  |  |  | 0.23 (0.769)
  Calcium, Day 2,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Calcium, Day 2,n=12,6,5,9,9,6 | -0.025 (0.0645) | -0.027 (0.0615) | -0.004 (0.0865) | -0.049 (0.0736) | 0.016 (0.1207) | 0.043 (0.0480)
  Calcium, Day 3,n=12,6,6,9,9,6 | 0.008 (0.0833) | -0.033 (0.1009) | 0.027 (0.1041) | -0.011 (0.0756) | -0.022 (0.1012) | 0.070 (0.0415)
  Calcium, Day 4,n=12,6,6,9,9,6 | 0.012 (0.0658) | -0.017 (0.0612) | 0.017 (0.0794) | -0.033 (0.0762) | -0.007 (0.0714) | 0.073 (0.0301)
  Calcium, Day 5,n=12,6,6,9,9,6 | -0.023 (0.0738) | -0.050 (0.0846) | 0.003 (0.0942) | -0.040 (0.0640) | -0.031 (0.0933) | 0.043 (0.0843)
  Calcium, Week 1,n=11,6,6,9,9,5: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 5
  Calcium, Week 1,n=11,6,6,9,9,5 | -0.009 (0.0745) | -0.047 (0.0723) | 0.017 (0.0916) | -0.044 (0.0847) | -0.029 (0.0657) | -0.040 (0.0663)
  Calcium, Week 2,n=12,6,6,9,9,6 | -0.007 (0.0634) | -0.013 (0.0547) | -0.033 (0.0855) | -0.002 (0.0863) | 0.062 (0.0771) | 0.013 (0.0163)
  Calcium, Week 4,n=12,6,6,9,9,6 | -0.040 (0.0615) | -0.027 (0.0766) | -0.013 (0.1198) | -0.031 (0.0729) | 0.022 (0.0977) | 0.033 (0.0301)
  Calcium, Week 8,n=12,6,6,9,9,6 | 0.000 (0.0621) | -0.007 (0.1171) | -0.003 (0.0898) | -0.024 (0.0767) | 0.031 (0.0906) | -0.003 (0.0612)
  Calcium, Week 12,n=12,6,6,9,9,6 | -0.017 (0.0489) | -0.060 (0.0657) | -0.003 (0.1274) | -0.020 (0.0755) | 0.036 (0.0581) | -0.003 (0.0794)
  Calcium, Week 18,n=12,6,6,9,9,6 | 0.003 (0.0918) | -0.013 (0.0826) | -0.033 (0.0845) | 0.007 (0.0860) | 0.031 (0.0801) | 0.010 (0.0690)
  Calcium, Week 24,n=12,6,6,9,9,6 | -0.035 (0.0452) | -0.053 (0.0677) | 0.007 (0.0864) | -0.016 (0.0942) | 0.022 (0.1218) | 0.027 (0.0797)
  Calcium, Week 26,n=12,6,6,9,9,6 | -0.018 (0.0731) | -0.067 (0.0532) | -0.017 (0.1255) | -0.056 (0.0260) | 0.013 (0.0529) | -0.010 (0.0767)
  Calcium, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Calcium, Week 32,n=6,6,6,0,0,6 | -0.020 (0.1020) | 0.027 (0.0776) | 0.020 (0.0867) |  |  | 0.010 (0.0724)
  Calcium, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Calcium, Week 36,n=6,0,0,9,9,0 | 0.000 (0.0607) |  |  | -0.013 (0.0624) | 0.029 (0.0813) |
  Calcium, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Calcium, Week 40,n=2,0,0,0,0,6 | 0.000 (0.1131) |  |  |  |  | 0.043 (0.0774)
  Potassium, Day 2,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Potassium, Day 2,n=12,6,5,9,9,6 | -0.03 (0.230) | 0.02 (0.179) | 0.44 (0.365) | 0.06 (0.397) | 0.18 (0.307) | 0.17 (0.234)
  Potassium, Day 3,n=12,6,6,9,9,6 | -0.07 (0.290) | 0.03 (0.258) | 0.02 (0.204) | 0.14 (0.332) | 0.01 (0.136) | 0.12 (0.194)
  Potassium, Day 4,n=12,6,6,9,9,6 | 0.13 (0.196) | 0.05 (0.472) | 0.08 (0.232) | 0.03 (0.218) | 0.06 (0.246) | 0.27 (0.163)
  Potassium, Day 5,n=12,6,6,9,9,6 | 0.11 (0.303) | 0.10 (0.276) | 0.00 (0.126) | 0.11 (0.267) | 0.04 (0.207) | 0.15 (0.217)
  Potassium, Week 1,n=11,6,6,9,9,5: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 5
  Potassium, Week 1,n=11,6,6,9,9,5 | -0.02 (0.340) | 0.05 (0.451) | 0.18 (0.194) | 0.22 (0.342) | 0.07 (0.300) | 0.00 (0.200)
  Potassium, Week 2,n=12,6,6,9,9,6 | 0.00 (0.316) | 0.05 (0.315) | 0.20 (0.341) | -0.04 (0.201) | 0.09 (0.352) | 0.02 (0.299)
  Potassium, Week 4,n=12,6,6,9,9,6 | 0.00 (0.276) | -0.07 (0.372) | 0.27 (0.344) | -0.04 (0.283) | 0.11 (0.196) | 0.00 (0.276)
  Potassium, Week 8,n=12,6,6,9,9,6 | 0.18 (0.234) | 0.00 (0.352) | 0.12 (0.117) | 0.00 (0.269) | 0.14 (0.207) | -0.05 (0.207)
  Potassium, Week 12,n=12,6,6,9,9,6 | -0.02 (0.383) | -0.02 (0.387) | 0.12 (0.331) | 0.00 (0.278) | 0.04 (0.213) | 0.03 (0.273)
  Potassium, Week 18,n=12,6,6,9,9,6 | -0.02 (0.343) | 0.00 (0.329) | 0.07 (0.234) | 0.03 (0.287) | 0.13 (0.308) | 0.02 (0.293)
  Potassium, Week 24,n=12,6,6,9,9,6 | -0.03 (0.458) | -0.02 (0.397) | 0.03 (0.234) | 0.12 (0.291) | -0.04 (0.260) | 0.07 (0.288)
  Potassium, Week 26,n=12,6,6,9,9,6 | -0.13 (0.360) | -0.03 (0.480) | 0.00 (0.179) | -0.01 (0.280) | 0.07 (0.235) | 0.07 (0.327)
  Potassium, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Potassium, Week 32,n=6,6,6,0,0,6 | -0.15 (0.476) | 0.03 (0.242) | 0.12 (0.223) |  |  | 0.12 (0.147)
  Potassium, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Potassium, Week 36,n=6,0,0,9,9,0 | 0.07 (0.121) |  |  | 0.08 (0.311) | 0.09 (0.215) |
  Potassium Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Potassium Week 40,n=2,0,0,0,0,6 | -0.35 (0.495) |  |  |  |  | 0.13 (0.356)
  Sodium, Day 2,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Sodium, Day 2,n=12,6,5,9,9,6 | 0.8 (2.14) | 0.0 (1.90) | 0.0 (1.58) | -0.3 (1.94) | 0.9 (1.76) | 1.8 (1.72)
  Sodium, Day 3,n=12,6,6,9,9,6 | 1.2 (1.75) | 0.0 (0.89) | 0.3 (1.21) | 0.4 (1.33) | 0.9 (1.96) | 2.0 (1.55)
  Sodium, Day 4,n=12,6,6,9,9,6 | 1.1 (1.93) | 0.2 (1.60) | 0.0 (2.19) | -0.8 (2.11) | 0.3 (1.32) | 1.3 (1.86)
  Sodium, Day 5,n=12,6,6,9,9,6 | 1.3 (1.66) | 1.7 (1.51) | -1.3 (1.86) | -0.2 (2.22) | 0.8 (2.05) | 1.7 (1.75)
  Sodium, Week 1,n=11,6,6,9,9,5: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 5
  Sodium, Week 1,n=11,6,6,9,9,5 | 0.8 (2.14) | 0.8 (2.32) | -1.7 (1.03) | 0.1 (1.45) | -0.1 (1.69) | 0.4 (2.19)
  Sodium, Week 2,n=12,6,6,9,9,6 | 0.1 (1.51) | 1.0 (1.26) | -0.7 (1.51) | 0.0 (1.32) | -0.3 (1.66) | 1.0 (2.28)
  Sodium, Week 4,n=12,6,6,9,9,6 | 0.0 (2.04) | 1.0 (1.41) | -1.2 (0.98) | -1.2 (1.30) | -0.6 (1.67) | 1.0 (1.41)
  Sodium, Week 8,n=12,6,6,9,9,6 | 0.1 (1.93) | 0.0 (2.53) | -0.5 (1.52) | -0.7 (1.94) | -1.1 (1.05) | 1.5 (3.45)
  Sodium, Week 12,n=12,6,6,9,9,6 | 0.0 (2.00) | 1.0 (1.26) | -0.8 (1.47) | -0.2 (1.56) | -0.3 (1.22) | 1.3 (2.25)
  Sodium, Week 18,n=12,6,6,9,9,6 | 0.1 (1.51) | -0.7 (2.25) | -1.0 (1.10) | -0.7 (1.22) | 0.0 (1.66) | 0.8 (1.60)
  Sodium, Week 24,n=12,6,6,9,9,6 | 0.3 (2.02) | -0.2 (1.60) | -1.5 (1.22) | -0.9 (2.37) | 0.2 (1.64) | 1.2 (1.72)
  Sodium, Week 26,n=12,6,6,9,9,6 | 0.2 (1.40) | 0.0 (1.90) | -0.7 (2.88) | -1.1 (2.15) | -1.1 (1.54) | 1.7 (1.97)
  Sodium, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Sodium, Week 32,n=6,6,6,0,0,6 | 0.3 (2.25) | 0.5 (3.56) | -1.8 (1.17) |  |  | 0.7 (2.07)
  Sodium, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Sodium, Week 36,n=6,0,0,9,9,0 | -0.3 (2.66) |  |  | -0.9 (1.90) | -1.3 (1.00) |
  Sodium, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Sodium, Week 40,n=2,0,0,0,0,6 | 0.5 (2.12) |  |  |  |  | 0.0 (1.90)
  Magnesium, Day 2,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  Magnesium, Day 2,n=12,6,5,9,9,6 | -0.020 (0.0467) | -0.037 (0.0585) | 0.008 (0.0642) | 0.000 (0.0361) | -0.036 (0.0623) | -0.020 (0.0310)
  Magnesium, Day 3,n=12,6,6,9,9,6 | -0.012 (0.0542) | -0.043 (0.0388) | -0.003 (0.0709) | 0.007 (0.0283) | -0.064 (0.0564) | -0.037 (0.0427)
  Magnesium, Day 4,n=12,6,6,9,9,6 | -0.013 (0.0750) | -0.020 (0.0310) | -0.007 (0.0575) | -0.007 (0.0283) | -0.060 (0.0490) | -0.047 (0.0628)
  Magnesium, Day 5,n=12,6,6,9,9,6 | -0.017 (0.0545) | -0.047 (0.0745) | -0.033 (0.0413) | 0.007 (0.0283) | -0.036 (0.0536) | -0.020 (0.0632)
  Magnesium, Week 1,n=11,6,6,9,9,5: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 5
  Magnesium, Week 1,n=11,6,6,9,9,5 | -0.004 (0.0427) | -0.003 (0.0638) | 0.017 (0.0480) | -0.007 (0.0520) | -0.040 (0.0346) | -0.032 (0.0460)
  Magnesium, Week 2,n=12,6,6,9,9,6 | 0.005 (0.0410) | -0.003 (0.0513) | 0.033 (0.0484) | 0.018 (0.0570) | -0.036 (0.0445) | -0.027 (0.0501)
  Magnesium, Week 4,n=12,6,6,9,9,6 | 0.007 (0.0345) | -0.033 (0.0589) | 0.000 (0.0456) | 0.007 (0.0346) | -0.027 (0.0529) | -0.017 (0.0408)
  Magnesium, Week 8,n=12,6,6,9,9,6 | -0.003 (0.0608) | -0.027 (0.0501) | -0.007 (0.0484) | 0.016 (0.0240) | -0.018 (0.0338) | -0.003 (0.0585)
  Magnesium, Week 12,n=12,6,6,9,9,6 | -0.013 (0.0492) | -0.043 (0.0686) | 0.000 (0.0551) | 0.011 (0.0448) | -0.011 (0.0501) | 0.000 (0.0456)
  Magnesium, Week 18,n=12,6,6,9,9,6 | 0.017 (0.0525) | -0.030 (0.0576) | 0.000 (0.0456) | 0.000 (0.0566) | -0.036 (0.0773) | 0.000 (0.0551)
  Magnesium, Week 24,n=12,6,6,9,9,6 | 0.008 (0.0422) | -0.023 (0.0585) | -0.017 (0.0686) | 0.000 (0.0424) | -0.047 (0.0557) | -0.003 (0.0320)
  Magnesium, Week 26,n=12,6,6,9,9,6 | 0.002 (0.0542) | -0.057 (0.0320) | -0.017 (0.0463) | 0.000 (0.0469) | -0.036 (0.0477) | -0.027 (0.0432)
  Magnesium, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  Magnesium, Week 32,n=6,6,6,0,0,6 | -0.010 (0.0245) | -0.023 (0.0497) | 0.017 (0.0480) |  |  | -0.027 (0.0301)
  Magnesium Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  Magnesium Week 36,n=6,0,0,9,9,0 | -0.013 (0.0532) |  |  | 0.004 (0.0133) | -0.013 (0.0447) |
  Magnesium, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  Magnesium, Week 40,n=2,0,0,0,0,6 | 0.030 (0.0424) |  |  |  |  | -0.030 (0.0329)
  BUN, Day 2,n=12,6,5,9,9,6: number analyzed (Participants) | 12 | 6 | 5 | 9 | 9 | 6
  BUN, Day 2,n=12,6,5,9,9,6 | -0.83 (1.135) | -0.17 (0.408) | 0.20 (1.304) | -0.67 (0.791) | -0.28 (0.833) | -1.25 (1.084)
  BUN, Day 3,n=12,6,6,9,9,6 | -0.79 (1.373) | 0.00 (0.316) | -0.17 (0.931) | -0.72 (0.833) | -0.28 (0.755) | -1.17 (1.402)
  BUN, Day 4,n=12,6,6,9,9,6 | -0.75 (1.357) | -0.25 (0.274) | -0.33 (1.169) | -0.61 (0.928) | 0.00 (0.707) | -0.50 (1.673)
  BUN, Day 5,n=12,6,6,9,9,6 | -0.71 (1.339) | -0.33 (0.816) | 0.67 (1.169) | -0.61 (0.961) | -0.17 (0.968) | -0.67 (1.602)
  BUN, Week 1,n=11,6,6,9,9,5: number analyzed (Participants) | 11 | 6 | 6 | 9 | 9 | 5
  BUN, Week 1,n=11,6,6,9,9,5 | -0.45 (1.150) | -0.50 (1.183) | 0.50 (1.581) | -0.44 (1.014) | 0.11 (0.782) | -1.10 (1.084)
  BUN, Week 2,n=12,6,6,9,9,6 | -0.33 (1.267) | -0.75 (1.037) | 0.33 (1.780) | 0.06 (0.726) | -0.17 (0.612) | -0.33 (1.080)
  BUN, Week 4,n=12,6,6,9,9,6 | -0.25 (1.098) | -0.75 (0.524) | 0.75 (0.822) | 0.22 (0.972) | 0.17 (1.225) | -0.08 (1.114)
  BUN, Week 8,n=12,6,6,9,9,6 | -0.75 (0.989) | -0.17 (1.033) | 1.17 (1.252) | 0.06 (1.074) | 0.28 (1.093) | -0.58 (1.158)
  BUN, Week 12,n=12,6,6,9,9,6 | -0.75 (1.323) | 0.17 (0.983) | 0.17 (0.816) | -0.06 (0.527) | 0.06 (0.682) | 0.25 (1.037)
  BUN, Week 18,n=12,6,6,9,9,6 | -1.08 (1.505) | 0.50 (1.414) | 0.58 (1.068) | 0.39 (1.516) | 0.00 (0.866) | -0.33 (0.983)
  BUN, Week 24,n=12,6,6,9,9,6 | -0.79 (1.389) | -0.17 (0.876) | 1.42 (1.594) | 0.11 (1.453) | 0.33 (1.146) | 0.17 (0.683)
  BUN, Week 26,n=12,6,6,9,9,6 | -0.38 (1.069) | -0.33 (0.983) | 0.83 (1.366) | -0.17 (1.000) | 0.22 (0.755) | 0.08 (1.068)
  BUN, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  BUN, Week 32,n=6,6,6,0,0,6 | -1.00 (0.949) | -0.33 (0.683) | 0.75 (1.405) |  |  | -0.08 (0.801)
  BUN, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  BUN, Week 36,n=6,0,0,9,9,0 | -0.58 (1.855) |  |  | -0.72 (1.034) | 0.28 (1.228) |
  BUN, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  BUN, Week 40,n=2,0,0,0,0,6 | -1.00 (0.000) |  |  |  |  | -0.42 (1.201)

57. Primary Outcome: Number of Participants With Presence of Ketones, Glucose, Occult Blood, and Protein
Description: Urine samples were collected to analyze presence of ketones, occult blood, glucose, and protein in urine. In this dipstick test, the level of occult blood, glucose, ketones and urine protein in urine samples were recorded as negative, trace, 1+ and 2+ indicating proportional concentrations in urine. Only categories with abnormal significant values have been presented.
Time Frame: Baseline and at Days 2, 3, 4 and 5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32, 36 and 40
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Participants
  Occult blood, Trace,Week 4,n=2,1,1,5,0,1: number analyzed (Participants) | 2 | 1 | 1 | 5 | 0 | 1
  Occult blood, Trace,Week 4,n=2,1,1,5,0,1 | 1 | 0 | 0 | 0 |  | 0
  Urine Ketone, Trace,Day 2,n=1,2,0,2,0,0: number analyzed (Participants) | 1 | 2 | 0 | 2 | 0 | 0
  Urine Ketone, Trace,Day 2,n=1,2,0,2,0,0 | 1 | 0 |  | 0 |  |
  Urine Ketone, Trace, Day 4,n=0,0,1,1,0,0: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 0
  Urine Ketone, Trace, Day 4,n=0,0,1,1,0,0 |  |  | 1 | 0 |  |
  Urine Ketone, Trace, Day 5,n=2,0,0,2,1,0: number analyzed (Participants) | 2 | 0 | 0 | 2 | 1 | 0
  Urine Ketone, Trace, Day 5,n=2,0,0,2,1,0 | 1 |  |  | 0 | 0 |
  Urine Ketone, Trace, Week 1,n=2,1,1,3,0,0: number analyzed (Participants) | 2 | 1 | 1 | 3 | 0 | 0
  Urine Ketone, Trace, Week 1,n=2,1,1,3,0,0 | 1 | 0 | 1 | 0 |  |
  Urine Ketone, Trace, Week 2,n=1,0,0,3,1,0: number analyzed (Participants) | 1 | 0 | 0 | 3 | 1 | 0
  Urine Ketone, Trace, Week 2,n=1,0,0,3,1,0 | 1 |  |  | 1 | 0 |
  Urine Ketone, Trace, Week 4,n=2,1,1,5,0,0: number analyzed (Participants) | 2 | 1 | 1 | 5 | 0 | 0
  Urine Ketone, Trace, Week 4,n=2,1,1,5,0,0 | 1 | 0 | 1 | 0 |  |
  Urine Ketone, Trace, Week 18,n=2,1,0,1,0,0: number analyzed (Participants) | 2 | 1 | 0 | 1 | 0 | 0
  Urine Ketone, Trace, Week 18,n=2,1,0,1,0,0 | 1 | 0 | 0 | 0 |  |
  Urine Ketone, Trace, Week 24,n=1,1,0,4,0,0: number analyzed (Participants) | 1 | 1 | 0 | 4 | 0 | 0
  Urine Ketone, Trace, Week 24,n=1,1,0,4,0,0 | 1 | 0 | 0 | 0 |  |
  Urine Ketone, Trace, Week 26,n=0,0,0,2,0,0: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0
  Urine Ketone, Trace, Week 26,n=0,0,0,2,0,0 |  |  |  | 1 |  |
  Urine Ketone, Trace,Week 32,n=1,0,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Urine Ketone, Trace,Week 32,n=1,0,0,0,0,0 | 1 |  |  |  |  |
  Urine Ketone, 1+, Week 40,n=0,0,0,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Urine Ketone, 1+, Week 40,n=0,0,0,0,0,1 |  |  |  |  |  | 1
  Urine Protein, 2+, Week 4,n=2,1,1,5,0,1: number analyzed (Participants) | 2 | 1 | 1 | 5 | 0 | 1
  Urine Protein, 2+, Week 4,n=2,1,1,5,0,1 | 1 | 0 | 0 | 0 |  | 0
  Urine Protein, Trace, Week 8,n=1,0,0,2,0,0: number analyzed (Participants) | 1 | 0 | 0 | 2 | 0 | 0
  Urine Protein, Trace, Week 8,n=1,0,0,2,0,0 | 1 |  |  | 0 |  |
  Urine Protein, Trace, Week 18,n=2,1,0,1,0,0: number analyzed (Participants) | 2 | 1 | 0 | 1 | 0 | 0
  Urine Protein, Trace, Week 18,n=2,1,0,1,0,0 | 1 | 0 |  | 0 |  |

58. Primary Outcome: Urine Potential of Hydrogen (pH) Analysis by Dipstick Method
Description: Urinary pH measurement is a routine part of urinalysis. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0).
Time Frame: Days 2, 3, 4 and 5, Weeks 1, 2, 4, 8, 12, 18, 24, 26, 32, 36 and 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 3 | 1 | 1 | 5 | 1 | 1
pH
  Day 2,n=1,1,0,2,0,0: number analyzed (Participants) | 1 | 1 | 0 | 2 | 0 | 0
  Day 2,n=1,1,0,2,0,0 | 5.00 (NA) — NA indicates that standard deviation could not be calculated for a single data point. | 7.00 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |  | 6.50 (1.414) |  |
  Day 3,n=3,0,0,1,0,0: number analyzed (Participants) | 3 | 0 | 0 | 1 | 0 | 0
  Day 3,n=3,0,0,1,0,0 | 6.00 (0.500) |  |  | 5.00 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |  |
  Day 4,n=0,0,1,1,0,0: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 0
  Day 4,n=0,0,1,1,0,0 |  |  | 6.50 (NA) — NA indicates that standard deviation could not be calculated for a single data point. | 5.00 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |  |
  Day 5,n=2,0,0,2,1,0: number analyzed (Participants) | 2 | 0 | 0 | 2 | 1 | 0
  Day 5,n=2,0,0,2,1,0 | 5.50 (0.707) |  |  | 5.75 (1.061) | 5.50 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |
  Week 1,n=2,1,1,3,0,0: number analyzed (Participants) | 2 | 1 | 1 | 3 | 0 | 0
  Week 1,n=2,1,1,3,0,0 | 5.50 (0.000) | 7.00 (NA) — NA indicates that standard deviation could not be calculated for a single data point. | 6.00 (NA) — NA indicates that standard deviation could not be calculated for a single data point. | 5.50 (0.500) |  |
  Week 2,n=1,0,0,4,1,0: number analyzed (Participants) | 1 | 0 | 0 | 4 | 1 | 0
  Week 2,n=1,0,0,4,1,0 | 5.50 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |  |  | 5.63 (0.479) | 8.50 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |
  Week 4,n=3,1,1,5,0,1: number analyzed (Participants) | 3 | 1 | 1 | 5 | 0 | 1
  Week 4,n=3,1,1,5,0,1 | 6.50 (0.866) | 8.00 (NA) — NA indicates that standard deviation could not be calculated for a single data point. | 5.50 (NA) — NA indicates that standard deviation could not be calculated for a single data point. | 6.00 (0.707) |  | 5.00 (NA) — NA indicates that standard deviation could not be calculated for a single data point.
  Week 8,n=1,0,0,2,0,0: number analyzed (Participants) | 1 | 0 | 0 | 2 | 0 | 0
  Week 8,n=1,0,0,2,0,0 | 5.50 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |  |  | 5.50 (0.000) |  |
  Week 12,n=0,1,0,1,0,0: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 0
  Week 12,n=0,1,0,1,0,0 |  | 6.50 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |  | 5.00 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |  |
  Week 18,n=3,1,0,1,0,0: number analyzed (Participants) | 3 | 1 | 0 | 1 | 0 | 0
  Week 18,n=3,1,0,1,0,0 | 5.67 (0.577) | 7.00 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |  | 5.00 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |  |
  Week 24,n=1,1,0,4,0,0: number analyzed (Participants) | 1 | 1 | 0 | 4 | 0 | 0
  Week 24,n=1,1,0,4,0,0 | 6.00 (NA) — NA indicates that standard deviation could not be calculated for a single data point. | 6.50 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |  | 5.38 (0.479) |  |
  Week 26,n=0,0,0,2,0,0: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0
  Week 26,n=0,0,0,2,0,0 |  |  |  | 5.50 (0.000) |  |
  Week 32,n=1,0,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Week 32,n=1,0,0,0,0,0 | 7.50 (NA) — NA indicates that standard deviation could not be calculated for a single data point. |  |  |  |  |
  Week 36,n=0,0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Week 40,n=0,0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

59. Primary Outcome: Absolute Values of Complement (C)3 and C4
Description: Blood samples were collected at indicated timepoints for analysis for complement (C3 and C4). Baseline was defined as latest pre-dose assessment with a non-missing value.
Time Frame: Baseline and at Days 2, 3, 4 and 5; Weeks 2, 4, 8, 12, 18, 24, 26, 32, 36 and 40
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Grams per liter
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
Number analyzed (Participants) | 12 | 6 | 6 | 9 | 9 | 6
Grams per liter
  C3, Baseline,n=12,6,6,9,9,6 | 1.149 [1.061 to 1.243] | 1.182 [0.995 to 1.404] | 1.086 [0.941 to 1.254] | 1.074 [0.982 to 1.175] | 1.137 [1.013 to 1.277] | 1.254 [1.122 to 1.402]
  C3, Day 2,n=12,6,6,9,9,6 | 1.13 [1.042 to 1.225] | 1.27 [1.051 to 1.535] | 1.16 [0.940 to 1.433] | 1.114 [1.018 to 1.219] | 1.188 [1.053 to 1.341] | 1.286 [1.182 to 1.400]
  C3, Day 3,n=12,6,6,9,9,6 | 1.187 [1.063 to 1.325] | 1.244 [1.029 to 1.503] | 1.236 [1.011 to 1.511] | 1.142 [1.037 to 1.258] | 1.157 [1.038 to 1.290] | 1.322 [1.197 to 1.460]
  C3, Day 4,n=12,6,6,9,9,6 | 1.17 [1.051 to 1.302] | 1.284 [1.023 to 1.611] | 1.181 [1.016 to 1.374] | 1.144 [1.051 to 1.245] | 1.165 [1.038 to 1.307] | 1.316 [1.189 to 1.458]
  C3, Day 5,n=12,6,6,9,9,6 | 1.136 [1.011 to 1.277] | 1.122 [0.993 to 1.268] | 1.092 [0.909 to 1.311] | 1.113 [1.011 to 1.226] | 1.165 [1.026 to 1.323] | 1.305 [1.159 to 1.469]
  C3, Week 2,n=12,6,6,9,9,6 | 1.136 [1.062 to 1.215] | 1.147 [0.986 to 1.333] | 1.02 [0.841 to 1.238] | 1.139 [1.045 to 1.241] | 1.174 [1.039 to 1.327] | 1.28 [1.136 to 1.442]
  C3, Week 4,n=12,6,6,9,9,6 | 1.114 [1.043 to 1.191] | 1.05 [0.873 to 1.262] | 1.111 [0.900 to 1.370] | 1.07 [0.957 to 1.197] | 1.148 [1.019 to 1.293] | 1.22 [1.085 to 1.372]
  C3, Week 8,n=12,6,6,9,9,6 | 1.224 [1.150 to 1.303] | 1.226 [1.115 to 1.347] | 1.097 [0.875 to 1.376] | 1.117 [0.993 to 1.257] | 1.167 [1.085 to 1.254] | 1.34 [1.191 to 1.506]
  C3, Week 12,n=12,6,6,9,9,6 | 1.117 [1.011 to 1.234] | 1.033 [0.935 to 1.141] | 1.124 [0.947 to 1.334] | 1.147 [1.050 to 1.254] | 1.211 [1.065 to 1.377] | 1.28 [1.117 to 1.465]
  C3, Week 18,n=12,6,6,9,9,6 | 1.173 [1.065 to 1.291] | 1.215 [0.984 to 1.500] | 1.124 [0.922 to 1.370] | 1.184 [1.045 to 1.342] | 1.231 [1.119 to 1.353] | 1.283 [1.158 to 1.422]
  C3, Week 24,n=12,6,6,8,9,6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 9 | 6
  C3, Week 24,n=12,6,6,8,9,6 | 1.15 [1.067 to 1.238] | 1.136 [1.031 to 1.252] | 1.171 [1.029 to 1.332] | 1.157 [1.019 to 1.312] | 1.243 [1.107 to 1.395] | 1.222 [1.100 to 1.356]
  C3, Week 26,n=12,6,6,9,9,6 | 1.204 [1.106 to 1.311] | 0.927 [0.450 to 1.910] | 1.142 [0.963 to 1.355] | 1.156 [1.070 to 1.249] | 1.222 [1.081 to 1.381] | 1.298 [1.123 to 1.501]
  C3, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  C3, Week 32,n=6,6,6,0,0,6 | 1.173 [0.985 to 1.398] | 1.243 [1.137 to 1.358] | 1.231 [1.016 to 1.491] |  |  | 1.204 [1.116 to 1.299]
  C3, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  C3, Week 36,n=6,0,0,9,9,0 | 1.243 [1.107 to 1.397] |  |  | 1.188 [1.085 to 1.301] | 1.236 [1.106 to 1.382] |
  C3, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  C3, Week 40,n=2,0,0,0,0,6 | 1.181 [NA to NA] — NA indicates not available as 95% Confidence Interval (CI) was only available when at least 3 participants contribute to the statistics |  |  |  |  | 1.231 [1.069 to 1.417]
  C4, Baseline,n=12,6,6,9,9,6 | 0.2576 [0.2108 to 0.3147] | 0.2061 [0.1653 to 0.2570] | 0.1919 [0.1337 to 0.2755] | 0.2144 [0.1727 to 0.2663] | 0.1939 [0.1496 to 0.2512] | 0.215 [0.1859 to 0.2488]
  C4, Day 2,n=12,6,6,9,9,6 | 0.2525 [0.2037 to 0.3130] | 0.2161 [0.1832 to 0.2549] | 0.2061 [0.1469 to 0.2891] | 0.2133 [0.1784 to 0.2549] | 0.203 [0.1597 to 0.2581] | 0.22 [0.1832 to 0.2643]
  C4, Day 3,n=12,6,6,9,9,6 | 0.2647 [0.2068 to 0.3389] | 0.2038 [0.1685 to 0.2464] | 0.2212 [0.1464 to 0.3342] | 0.2142 [0.1759 to 0.2609] | 0.1962 [0.1514 to 0.2544] | 0.223 [0.1921 to 0.2589]
  C4, Day 4,n=12,6,6,9,9,6 | 0.253 [0.2013 to 0.3179] | 0.2303 [0.1918 to 0.2767] | 0.2006 [0.1416 to 0.2842] | 0.2128 [0.1766 to 0.2564] | 0.1935 [0.1472 to 0.2543] | 0.2188 [0.1867 to 0.2564]
  C4, Day 5,n=12,6,6,9,9,6 | 0.2497 [0.1929 to 0.3232] | 0.1892 [0.1572 to 0.2277] | 0.1866 [0.1327 to 0.2680] | 0.2073 [0.1685 to 0.2551] | 0.1943 [0.1492 to 0.2531] | 0.2163 [0.1869 to 0.2503]
  C4, Week 2,n=12,6,6,9,9,6 | 0.2555 [0.2028 to 0.3220] | 0.2108 [0.1768 to 0.2514] | 0.1781 [0.1172 to 0.2706] | 0.221 [0.1813 to 0.2695] | 0.2018 [0.1497 to 0.2720] | 0.2169 [0.1765 to 0.2664]
  C4, Week 4,n=12,6,6,9,9,6 | 0.2602 [0.2078 to 0.3258] | 0.1928 [0.1623 to 0.2290] | 0.189 [0.1292 to 0.2766] | 0.2063 [0.1636 to 0.2602] | 0.1872 [0.1419 to 0.2468] | 0.1929 [0.1733 to 0.2146]
  C4, Week 8,n=12,6,6,9,9,6 | 0.2738 [0.2186 to 0.3431] | 0.2547 [0.2010 to 0.3226] | 0.2045 [0.1315 to 0.3180] | 0.2009 [0.1654 to 0.2441] | 0.1901 [0.1542 to 0.2343] | 0.2231 [0.1778 to 0.2800]
  C4, Week 12,n=12,6,6,9,9,6 | 0.2413 [0.1901 to 0.3063] | 0.1862 [0.1567 to 0.2213] | 0.2034 [0.1307 to 0.3167] | 0.2114 [0.1723 to 0.2594] | 0.196 [0.1494 to 0.2572] | 0.2074 [0.1792 to 0.2400]
  C4, Week 18,n=12,6,6,9,9,6 | 0.261 [0.1992 to 0.3420] | 0.2266 [0.1873 to 0.2742] | 0.2025 [0.1322 to 0.3102] | 0.226 [0.1920 to 0.2660] | 0.1678 [0.1255 to 0.2245] | 0.216 [0.1740 to 0.2681]
  C4, Week 24,n=12,6,6,8,9,6: number analyzed (Participants) | 12 | 6 | 6 | 8 | 9 | 6
  C4, Week 24,n=12,6,6,8,9,6 | 0.2474 [0.1894 to 0.3232] | 0.2244 [0.1742 to 0.2890] | 0.197 [0.1324 to 0.2932] | 0.206 [0.1801 to 0.2357] | 0.1909 [0.1500 to 0.2430] | 0.2114 [0.1682 to 0.2658]
  C4, Week 26,n=12,6,6,9,9,6 | 0.2517 [0.1926 to 0.3291] | 0.202 [0.1319 to 0.3095] | 0.1939 [0.1291 to 0.2912] | 0.2115 [0.1704 to 0.2627] | 0.163 [0.1250 to 0.2126] | 0.226 [0.1887 to 0.2627]
  C4, Week 32,n=6,6,6,0,0,6: number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 6
  C4, Week 32,n=6,6,6,0,0,6 | 0.2772 [0.1617 to 0.4754] | 0.2401 [0.2003 to 0.2877] | 0.2007 [0.1297 to 0.3105] |  |  | 0.2051 [0.1808 to 0.2326]
  C4, Week 36,n=6,0,0,9,9,0: number analyzed (Participants) | 6 | 0 | 0 | 9 | 9 | 0
  C4, Week 36,n=6,0,0,9,9,0 | 0.2844 [0.2110 to 0.3834] |  |  | 0.2025 [0.1637 to 0.2504] | 0.206 [0.1626 to 0.2611] |
  C4, Week 40,n=2,0,0,0,0,6: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 6
  C4, Week 40,n=2,0,0,0,0,6 | 0.1699 [NA to NA] — NA indicates not available as 95% Confidence Interval (CI) was only available when at least 3 participants contribute to the statistics |  |  |  |  | 0.2134 [0.1766 to 0.2580]

ADVERSE EVENTS:
Time Frame: Non-serious AEs and SAEs were collected from the start of the study treatment (Day 1) up to Week 32 for GSK3511294 2 mg and 10 mg, up to Week 36 for GSK3511294 30 mg and GSK3511294 100 mg and up to Week 40 for GSK3511294 300 mg; and up to 40 weeks for placebo.
Description: Non-SAEs and SAEs were reported for the Safety Population. Within each cohort participants were assigned to active or placebo in a 3:1 ratio. A pooled placebo group was to be used as comparison group. An identical proportion of participants in pooled placebo group had same total duration of study as participants in each of the active dose groups
Arm/Group | Placebo | GSK3511294 2mg | GSK3511294 10mg | GSK3511294 30mg | GSK3511294 100mg | GSK3511294 300mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/9 | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/9 | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 11/12 | 2/6 | 6/6 | 8/9 | 9/9 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | GSK3511294 2mg (N=6) | GSK3511294 10mg (N=6) | GSK3511294 30mg (N=9) | GSK3511294 100mg (N=9) | GSK3511294 300mg (N=6)
Nasopharyngitis (Infections and infestations) | 2 (3) | 2 (4) | 1 (1) | 3 (3) | 5 (5) | 2 (2)
Rhinitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Root canal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral diarrhoea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 2 (4) | 3 (4) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Splinter (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental pulp disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 1 (4)
Allergy to animal (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peak expiratory flow rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (4)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental care (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site reaction (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hernia pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT03287310/SAP_000.pdf
  • Study Protocol (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT03287310/Prot_001.pdf